CLINICAL TRIAL: NCT01208662
Title: A Randomized, Phase III Study Comparing Conventional Dose Treatment Using a Combination of Lenalidomide, Bortezomib, and Dexamethasone (RVD) to High-Dose Treatment With Peripheral Stem Cell Transplant in the Initial Management of Myeloma in Patients Up to 65 Years of Age
Brief Title: Randomized Trial of Lenalidomide, Bortezomib, Dexamethasone vs High-Dose Treatment With SCT in MM Patients up to Age 65
Acronym: DFCI 10-106
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Paul Richardson, MD (Other)
Collaborators: Celgene Corporation (Industry); Millennium Pharmaceuticals, Inc. (Industry); Massachusetts General Hospital (Other); Cape Cod Hospital (Other); Beth Israel Deaconess Medical Center (Other); Emory University (Other); University of Michigan (Other); Fox Chase Cancer Center (Other); Memorial Sloan Kettering Cancer Center (Other); Fred Hutchinson Cancer Center (Other); Barbara Ann Karmanos Cancer Institute (Other); Duke University (Other); University of California, San Francisco (Other); University of Chicago (Other); M.D. Anderson Cancer Center (Other); UNC Lineberger Comprehensive Cancer Center (Other); Roswell Park Cancer Institute (Other); Stanford University (Other); University of Mississippi Medical Center (Other); Icahn School of Medicine at Mount Sinai (Other); Wake Forest University Health Sciences (Other); University of Arizona (Other); OHSU Knight Cancer Institute (Other); Eastern Maine Medical Center (Other); University of California, San Diego (Other); University of Alabama at Birmingham (Other); University of Pittsburgh Medical Center (Other); Ochsner Health System (Other); University of Texas Southwestern Medical Center (Other); State University of New York - Downstate Medical Center (Other); Newton-Wellesley Hospital (Other); Baylor College of Medicine (Other); City of Hope Medical Center (Other); University of Florida (Other); Northwell Health (Other); H. Lee Moffitt Cancer Center and Research Institute (Other); Vanderbilt University Medical Center (Other); Ohio State University (Other); Huntsman Cancer Institute (Other); Columbia University (Other)
Responsible Party: Sponsor-Investigator, Paul Richardson, MD, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-106
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Results first posted 2023-12-18 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: Lenalidomide; Bortezomib; Dexamethasone; Stem Cell Transplant; Myeloma; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Lenalidomide; Bortezomib; Dexamethasone; Calcium Dobesilate; Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RVD Alone (Experimental): All participants received one cycle of Lenalidomide (R), bortezomib (V) and dexamethasone (D) and then were randomized. All participants then received two additional RVD cycles, followed by stem-cell collection. RVD Alone participants received five additional RVD cycles. Maintenance in both arms comprised daily lenalidomide 10 mg, escalated to 15 mg if tolerated, until disease progression, unacceptable toxicity, or withdrawal from treatment or study. After finishing protocol-specified treatment, off-study salvage transplantation was recommended but not mandated for RVD Alone participants at relapse.
  RVD cycle duration=21 days R: 25 mg oral on days 1-14 V: 1.3 mg per square meter of body surface area IV or subcutaneous on days 1, 4, 8, and 11 D: 20 mg oral (cycles 1-3) or 10 mg (cycles 4-8) on days 1, 2, 4, 5, 8, 9, 11, and 12
  Interventions: Drug: Lenalidomide; Drug: Bortezomib; Drug: Dexamethasone
- RVD plus ASCT (Active Comparator): All participants received one cycle of Lenalidomide (R), bortezomib (V) and dexamethasone (d) and then were randomized. All participants then received two additional RVD cycles, followed by stem-cell collection. RVD plus autologous stem cell transplant (ASCT) participants received high-dose melphalan (200 mg/m2, adjusted for ideal body weight) ASCT and, upon recovery (~day 60), two additional RVD cycles. Maintenance in both arms comprised daily lenalidomide 10 mg, escalated to 15 mg if tolerated, until disease progression, unacceptable toxicity, or withdrawal from treatment or study.
  After finishing protocol-specified treatment, RVD plus ASCT participants could undergo a second transplant.
  RVD cycle duration=21 days R: 25 mg oral on days 1-14 V: 1.3 mg per square meter of body surface area IV or subcutaneous on days 1, 4, 8, and 11 D: 20 mg oral (cycles 1-3) or 10 mg (cycles 4-8) on days 1, 2, 4, 5, 8, 9, 11, and 12
  Interventions: Drug: Lenalidomide; Drug: Bortezomib; Drug: Dexamethasone; Procedure: Autologous Stem Cell Transplant

INTERVENTIONS:
Drug: Lenalidomide — oral administration
  Other Names: CC-5013
Drug: Bortezomib — intravenous or, following protocol amendment, subcutaneous administration
  Other Names: PS-341; Velcade
Drug: Dexamethasone — oral administration
  Dose of 20 mg/day for first 3 cycles. Dose of 10 mg/day for remaining cycles.
  Other Names: Decadron
Procedure: Autologous Stem Cell Transplant — Autologous refers to stem cells that are harvested from the participant to be a source of new blood cells after high-dose chemotherapy with melphalan.
  Other Names: Peripheral Blood Stem Cell (PBSC) Transplant
  Arms: RVD plus ASCT

SUMMARY:
In this research study, we are looking to explore the drug combination, lenalidomide, bortezomib and dexamethasone alone or when combined with autologous stem cell transplantation to see what side effects it may have and how well it works for treatment of newly diagnosed multiple myeloma. Specifically, the objective of this trial is to determine if, in the era of novel drugs, high dose therapy (HDT) is still necessary in the initial management of multiple myeloma in younger patients. In this study, HDT as compared to conventional dose treatment would be considered superior if it significantly prolongs progression-free survival by at least 9 months or more, recognizing that particular subgroups may benefit more compared to others.

DETAILED DESCRIPTION:
The drugs, lenalidomide, bortezomib, and dexamethasone, are approved by the FDA. They have not been approved in the combination for multiple myeloma or any other type of cancer. Bortezomib is currently approved by the FDA for the treatment of multiple myeloma. Lenalidomide is approved for use with dexamethasone for patients with multiple myeloma who have received at least one prior therapy and for the treatment of certain types of myelodysplastic syndrome (another type of cancer affecting the blood). Dexamethasone is commonly used, either alone, or in combination with other drugs, to treat multiple myeloma. Please note that Bortezomib and Lenalidomide are provided to patients participating in this trial at no charge. Melphalan and cyclophosphamide, the drugs used during stem cell collection and transplant, are also approved by the FDA. Melphalan is an FDA-approved chemotherapy for multiple myeloma and is used as a high-dose conditioning treatment prior to stem cell transplantation. Cyclophosphamide is used, either alone, or in combination with other drugs, to treat multiple myeloma. These drugs have been used in other multiple myeloma studies and information from those studies suggests that this combination of therapy may help to treat newly diagnosed multiple myeloma.

After screening procedures determine if a patient is eligible for this research study, the patient will be randomized into one of the study groups: lenalidomide, bortezomib and dexamethasone without autologous stem cell transplantation, followed by lenalidomide maintenance (Arm A) or lenalidomide, bortezomib and dexamethasone with autologous stem cell transplantation, followed by lenalidomide maintenance (Arm B). There is an equal chance of being placed in either group. Randomization was stratified by International Staging System (ISS) disease stage (I, II, or III) and cytogenetics (high-risk [presence of 17p deletion, t(4;14), or t(14;16) on fluorescence in-situ hybridization], standard-risk [absence of high-risk abnormalities], or undetermined [test failure]) assessed locally in a screening bone marrow sample, with positivity cut-offs per institutional standards.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Multiple Myeloma, according to the International Myeloma Foundation 2003 Diagnostic Criteria
* Documented symptomatic myeloma, with organ damage related to myeloma with laboratory assessments performed within 21 days of registration
* Myeloma that is measurable by either serum or urine evaluation of the monoclonal component or by assay of serum free light chains.
* ECOG performance status </= 2
* Negative HIV blood test
* Voluntary written informed consent

Exclusion Criteria:

* Pregnant or lactating female
* Prior systemic therapy for MM (localized radiotherapy allowed if at least 7 days before study entry, corticosteroids allowed if dose </= equivalent of 160 mg dexamethasone over 2 weeks)
* Primary amyloidosis (AL) or myeloma complicated by amylosis
* Receiving any other investigational agents
* Known brain metastases
* Poor tolerability or allergy to any of the study drugs or compounds of similar composition
* Platelet count <50,000/mm3, within 21 days of registration
* ANC <1,000 cells/mm3, within 21 days of registration
* Hemoglobin <8 g/dL, within 21 days of registration
* Hepatic impairment (>/= 1.5 x institutional ULN or AST (SGOT), ALT (SGPT), or alkaline phosphatase >2 x ULN). Patients with benign hyperbilirubinemia are eligible.
* Renal insufficiency (serum creatinine >2.0 mg/dl or creatinine clearance <50 ml/min, within 21 days of registration)
* Respiratory compromise (DLCO < 50%)
* Clinical signs of heart or coronary failure or LVEF < 40%. Myocardial infarction within 6 months prior to enrollment, NYHA Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conductive system abnormalities
* Intercurrent illness including, but not limited to ongoing or active severe infection, known infection with hepatitis B or C virus, poorly controlled diabetes, severe uncontrolled psychiatric disorder or psychiatric illness/social situations that would limit compliance with study requirements
* Previous history of another malignant condition except for basal cell carcinoma and stage I cervical cancer. If malignancy was experienced more than 2 years ago and confirmed as cured, these participants may be considered for the study on case by case basis with PI discussion.
* Inability to comply with an anti-thrombotic treatment regimen
* Peripheral neuropathy >/= Grade 2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 729 (Actual)
Dates: Start 2010-09; Primary Completion 2022-02 (Actual); Study Completion 2026-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Paul G. Richardson, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (46):
- United States (46):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Comprehensive Cancer Center, Tucson, Arizona
  - City of Hope, Duarte, California
  - University of California at San Diego, La Jolla, California
  - University of California, San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - University of Chicago, Chicago, Illinois
  - Ochsner Foundation Clinic, New Orleans, Louisiana
  - Eastern Maine Medical Center, Brewer, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Cape Cod Healthcare, Hyannis, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - New Hampshire Oncology and Hematology, Concord, New Hampshire
  - New Hampshire Oncology and Hematology, Hooksett, New Hampshire
  - New Hampshire Oncology and Hematology, Laconia, New Hampshire
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore Long Island Jewish Health System, Lake Success, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Oregon Health and Sciences, Portland, Oregon
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Richardson PG, Jacobus SJ, Weller EA, Hassoun H, Lonial S, Raje NS, Medvedova E, McCarthy PL, Libby EN, Voorhees PM, Orlowski RZ, Anderson LD Jr, Zonder JA, Milner CP, Gasparetto C, Agha ME, Khan AM, Hurd DD, Gowin K, Kamble RT, Jagannath S, Nathwani N, Alsina M, Cornell RF, Hashmi H, Campagnaro EL, Andreescu AC, Gentile T, Liedtke M, Godby KN, Cohen AD, Openshaw TH, Pasquini MC, Giralt SA, Kaufman JL, Yee AJ, Scott E, Torka P, Foley A, Fulciniti M, Hebert K, Samur MK, Masone K, Maglio ME, Zeytoonjian AA, Nadeem O, Schlossman RL, Laubach JP, Paba-Prada C, Ghobrial IM, Perrot A, Moreau P, Avet-Loiseau H, Attal M, Anderson KC, Munshi NC; DETERMINATION Investigators. Triplet Therapy, Transplantation, and Maintenance until Progression in Myeloma. N Engl J Med. 2022 Jul 14;387(2):132-147. doi: 10.1056/NEJMoa2204925. Epub 2022 Jun 5. PMID 35660812
- [Derived] Parmar H, Vesole DH, Biran N. From VAD to VRD: Is Transplant Still Needed in the Upfront Setting of Myeloma? Cancer J. 2021 May-Jun 01;27(3):190-195. doi: 10.1097/PPO.0000000000000522. PMID 34549906

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 56 clinical sites in the U.S. from Oct 1, 2010 to January 30, 2018.
Groups:
- RVD Cycle 1 Only: Some participants started cycle 1 lenalidomide (R), bortezomib (V) and dexamethasone (D) therapy but were not randomized.
  RVD cycle duration=21 days R: 25 mg oral on days 1-14 V: 1.3 mg per square meter of body surface area IV or subcutaneous on days 1, 4, 8, and 11 D: 20 mg oral (cycles 1) on days 1, 2, 4, 5, 8, 9, 11, and 12
Period: Induction and Consolidation
Arm/Group | RVD Alone | RVD Plus ASCT | RVD Cycle 1 Only
Started | 357 | 365 | 7
Randomized (Participants were randomized after 1 cycle of therapy only if cycle 1 therapy was completed and/or participant did not withdraw.) | 357 | 365 | 0
Underwent Stem Cell Mobilization | 324 | 330 | 0
Completed | 291 | 289 | 0
Not Completed | 66 | 76 | 7
Not completed — Disease Progression | 23 | 13 | 0
Not completed — Adverse Event | 16 | 18 | 2
Not completed — MD or Participant Decision | 16 | 34 | 4
Not completed — Death | 1 | 3 | 1
Not completed — Discontinued for other reasons | 10 | 8 | 0
Period: Maintenance
Arm/Group | RVD Alone | RVD Plus ASCT | RVD Cycle 1 Only
Started | 291 | 289 | 0
Minimal Residual Disease (MRD) Evaluable at Maintenance Start (MRD evaluable subset represents participants with clonal sequence identified at baseline plus MRD assessment at start of maintenance.) | 108 | 90 | 0
Completed (Given maintenance treatment duration is not fixed, all participants are considered as 'Not Completed'.) | 0 | 0 | 0
Not Completed | 291 | 289 | 0
Not completed — Disease Progression | 156 | 102 | 0
Not completed — Adverse Event | 12 | 28 | 0
Not completed — MD or Participant Decision | 24 | 36 | 0
Not completed — Death | 0 | 3 | 0
Not completed — Discontinued for other reasons | 21 | 31 | 0
Not completed — Still on Treatment | 78 | 89 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- RVD Cycle 1 Only: Some participants started cycle 1 lenalidomide (R), bortezomib (V) and dexamethasone (D) therapy but were not randomized.
  RVD cycle duration=21 days R: 25 mg oral on days 1-14 V: 1.3 mg per square meter of body surface area IV or subcutaneous on days 1, 4, 8, and 11 D: 20 mg oral (cycles 1-3) or 10 mg (cycles 4-8) on days 1, 2, 4, 5, 8, 9, 11, and 12
- Total: Total of all reporting groups
Arm/Group | RVD Alone | RVD Plus ASCT | RVD Cycle 1 Only | Total
Number analyzed (Participants) | 357 | 365 | 7 | 729
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [25 to 66] | 55 [30 to 65] | 59 [55 to 65] | 56 [50 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155 | 150 | 3 | 308
  Male | 202 | 215 | 4 | 421
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 23 | 0 | 42
  Not Hispanic or Latino | 336 | 332 | 7 | 675
  Unknown or Not Reported | 2 | 10 | 0 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 268 | 272 | 5 | 545
  Black | 66 | 66 | 2 | 134
  Asian | 8 | 12 | 0 | 20
  Other | 9 | 9 | 0 | 18
  Unknown | 6 | 6 | 0 | 12
Region of Enrollment [Number; unit: participants]
  United States | 357 | 365 | 7 | 729
ISS Multiple Myeloma Stage [Count of Participants; unit: Participants] — The International Staging System (ISS) consists of three stages: stage I, serum beta 2-microglobulin level lower than 3.5 mg per liter and serum albumin level 3.5 g per deciliter or higher; stage II, neither stage I nor III; and stage III, serum beta 2-microglobulin level 5.5 mg per liter or higher. Higher stages indicate more severe disease. Population: ISS Multiple Myeloma staging data collected at randomization and therefore data was not collected for the seven participants who were not randomized.
  Participants
    I: number analyzed (Participants) | 357 | 365 | 0 | 722
    I | 178 | 184 |  | 362
    II: number analyzed (Participants) | 357 | 365 | 0 | 722
    II | 130 | 134 |  | 264
    III: number analyzed (Participants) | 357 | 365 | 0 | 722
    III | 49 | 47 |  | 96
Cytogenetic Risk Category [Count of Participants; unit: Participants] — Cytogenetic risk was based on FISH or karyotype analysis; patients who had a high-risk cytogenetic profile had at least one high-risk abnormality (t[4;14], t[14;16], or del17p). Patients with standard risk had no high-risk cytogenetic abnormalities. Population: Cytogenetic risk category data collected at randomization and therefore data was not collected for the seven participants who were not randomized.
  Participants
    High risk: number analyzed (Participants) | 357 | 365 | 0 | 722
    High risk | 66 | 66 |  | 132
    Standard risk: number analyzed (Participants) | 357 | 365 | 0 | 722
    Standard risk | 268 | 274 |  | 542
BMI [Count of Participants; unit: Participants] — The body-mass index (BMI) is the weight in kilograms divided by the square of the height in meters.
  Participants
    <25 | 80 | 81 | 1 | 162
    25 to <30 | 141 | 127 | 2 | 270
    >/= 30 | 136 | 157 | 4 | 297
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status: (PS0) Fully active, able to carry on all pre-disease performance without restriction (PS1) Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (PS2) Ambulatory and capable of all self-care but unable to carry out any work activities; Up and about >50% of waking hours.
  Participants
    0 | 153 | 164 | 4 | 321
    1 | 177 | 161 | 3 | 341
    2 | 27 | 39 | 0 | 66
    Unknown | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Median Progression-Free Survival (PFS)
Description: PFS was estimated using the Kaplan-Meier (KM) method and defined as time from randomization to the earlier of disease progression (PD) as determined by central review or death from any cause (events). Patients who started non-protocol therapy (NPT) were censored at the date of NPT initiation if available or date treatment ended if date of NPT was missing. Deaths occurring beyond 1 year from the date last known progression-free are not counted as events and censored at date of last disease evaluation. Patients who had not started NPT, progressed, or died were censored at the date of last disease evaluation. PD was based upon the International Myeloma Working Group (IMWG) uniform response criteria. [Kumar S, et al Lancet Oncol 2016;17(8):e328-e346].
Time Frame: On treatment, disease was assessed every cycle up to maintenance and every 3 cycles on maintenance. In long-term follow-up, disease was assessed every 2 months until PD or death. Median (maximum) PFS follow-up was 70 and 129 months.
Population: The analysis population is comprised of all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RVD Alone | RVD Plus ASCT
Number analyzed (Participants) | 357 | 365
months | 46.2 [38.1 to 53.7] | 67.5 [58.6 to NA] — 95% CI upper bound not estimable because data not mature enough. Specifically, with the follow-up observed as of data extraction, there were not enough events.
Statistical Analysis 1: Comparison: RVD Alone vs RVD Plus ASCT; Test type: Superiority; p < 0.001, Log Rank; Observed Stratified Log Rank Test (1-sided p-value); Hazard Ratio (HR) = 1.53, 95% CI 2-sided [1.23 to 1.91]

2. Secondary Outcome: Partial Response (PR) Rate
Description: The PR rate is the percentage of participants achieving PR or better on treatment and was evaluated based on the IMWG criteria. PR was defined as > 50% reduction of serum M-protein and reduction in 24-h urinary M-protein by > 90% or to < 200mg per 24 hours. If the serum and urine M-protein are unmeasurable, a > 50% decrease in the difference between involved and uninvolved free light chain levels is required in place of the M-protein criteria. If serum and urine M-protein are unmeasurable, and serum free light assay is also unmeasurable, >50% reduction in plasma cells is required in place of M-protein, provided baseline bone marrow plasma cell percentage was > 30%. In addition to the above listed criteria, if present at baseline, a > 50% reduction in the size of soft tissue plasmacytomas was also required. Exact (Clopper-Pearson) confidence limits of 98.2857% represents Bonferroni adjustment for 7 tests (1-0.05/7) per statistical analysis plan for key secondary outcomes.
Time Frame: Disease was assessed every cycle up to maintenance and every 3 cycles on maintenance. Median treatment duration (months) from randomization 28.2 (RVD Alone) and 36.1 (RVD plus ASCT). Maximum treatment duration was 133.5 months in this study cohort.
Population: The analysis population is comprised of all randomized participants.
Measure: Number (99.29% Confidence Interval); unit: percentage of participants
Arm/Group | RVD Alone | RVD Plus ASCT
Number analyzed (Participants) | 357 | 365
percentage of participants | 95 [91.0 to 97.5] | 97.5 [94.5 to 99.2]
Statistical Analysis 1: Comparison: RVD Alone vs RVD Plus ASCT; Exact (Clopper-Pearson) confidence limits of 98.2857% represents Bonferroni adjustment for 7 tests (1-0.05/7) per statistical analysis plan for key secondary outcomes; Test type: Superiority; p = 0.55, Fisher Exact

3. Secondary Outcome: Very Good Partial Response (VGPR) Rate
Description: The VGPR rate is the percentage of participants achieving VGPR or better on treatment and was evaluated based on IMWG criteria. VGPR was defined as serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level <100mg per 24 hours.
Time Frame: Disease was assessed every cycle up to maintenance and every 3 cycles on maintenance. Median treatment duration (months) from randomization 28.2 (RVD Alone) and 36.1 (RVD plus ASCT). Maximum treatment duration was 134 months in this study cohort.
Population: The analysis population is comprised of all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | RVD Alone | RVD Plus ASCT
Number analyzed (Participants) | 357 | 365
percentage of patients | 79.6 [73.3 to 85.0] | 82.7 [76.8 to 87.7]
Statistical Analysis 1: Comparison: RVD Alone vs RVD Plus ASCT; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.99, Fisher Exact

4. Secondary Outcome: Complete Response (CR) Rate
Description: The CR rate is the percentage of participants achieving CR or better on treatment and was evaluated based on IMWG criteria. CR was defined as the negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow. Confirmation with repeat bone marrow biopsy was not needed.
Time Frame: as for outcome 3
Population: The analysis population is comprised of all randomized patients.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | RVD Alone | RVD Plus ASCT
Number analyzed (Participants) | 357 | 365
percentage of patients | 42.0 [35.0 to 49.3] | 46.8 [39.8 to 54.0]
Statistical Analysis 1: Comparison: RVD Alone vs RVD Plus ASCT; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.99, Fisher Exact

5. Secondary Outcome: Median Duration of Response: Partial Response (DOR PR)
Description: DOR PR was estimated using the KM method and defined as the time from documented best response as CR to documented disease progression per IMWG criteria. Patients who have not progressed or died were censored at the date last known progression-free.
Time Frame: On treatment, disease was assessed every cycle up to maintenance and every 3 cycles on maintenance. In long-term follow-up, disease was assessed every 2 months until PD or death. Median (maximum) DOR PR follow-up was 62.9 and 122.9 months.
Population: The analysis population is comprised of all randomized participants who achieved PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RVD Alone | RVD Plus ASCT
Number analyzed (Participants) | 339 | 356
months | 38.9 [30.8 to 45.6] | 56.4 [47.4 to 75.8]

6. Secondary Outcome: 5-Year Time to Progression (TTP)
Description: TTP was estimated using the KM method and defined as time from randomization to time of documented IMWG disease progression or censoring time (time of last disease evaluation for those alive, time to death among those who died). Patients initiating non-protocol therapy prior to progression or death were censored at the date of non-protocol therapy in the TTP analysis. The 5-year TTP endpoint is a probability.
Time Frame: On treatment, disease was assessed every cycle up to maintenance and every 3 cycles on maintenance. In long-term follow-up, disease was assessed every 2 months until PD or death. Median TTP follow-up was 70 months. The probability estimate is at 5 years.
Population: The analysis population is comprised of all randomized participants.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | RVD Alone | RVD Plus ASCT
Number analyzed (Participants) | 357 | 365
percent probability | 41.6 [35.8 to 47.3] | 58.4 [52.2 to 64.2]
Statistical Analysis 1: Comparison: RVD Alone vs RVD Plus ASCT; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Log Rank; Stratified; Hazard Ratio (HR) = 1.66, 99.29% CI 2-sided [1.21 to 2.27]

7. Secondary Outcome: 5-Year Overall Survival (OS)
Description: OS was estimated using the KM method and defined as time from randomization to death due to any cause. Patients alive were censored at date last known alive. The 5-year OS endpoint is a probability.
Time Frame: In long-term follow-up, survival follow-up every 2 months until death. Median (maximum) OS follow-up was 76 and 129 months.The probability estimate is at 5 years.
Population: The analysis population is comprised of all randomized participants.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | RVD Alone | RVD Plus ASCT
Number analyzed (Participants) | 357 | 365
percent probability | 79.2 [74.3 to 83.3] | 80.7 [76.1 to 84.6]
Statistical Analysis 1: Comparison: RVD Alone vs RVD Plus ASCT; Test type: Superiority; p > 0.99, Log Rank; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.73 to 1.65]

8. Secondary Outcome: Grade 3 or Higher Treatment-Related Non-Hematologic Adverse Event (AE) Rate
Description: Safety was evaluated throughout trial treatment, including ASCT, and through 30 days after receipt of the last dose of a trial drug. Treatment attribution and grade were based on the NCI CTCAE v4. The Grade 3 or Higher Treatment-Related Non-Hematologic AE Rate is percentage of participants who experienced any grade 3-5 treatment-related (possible, probable or definite attribution) non-hematologic adverse event based on CTCAEv4 as reported on case report forms. The difference in the rate of all grade 3 or higher toxicities was compared between the two groups using Fisher's exact test.
Time Frame: AEs was assessed every cycle on treatment. Median treatment duration (months) from randomization 28.2 (RVD Alone) and 36.1 (RVD plus ASCT). Maximum treatment duration was 133.5 months in this study cohort.
Population: The analysis population comprised of all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RVD Alone | RVD Plus ASCT
Number analyzed (Participants) | 357 | 365
percentage of participants | 78.2 [73.5 to 82.3] | 94.2 [91.3 to 96.4]

9. Secondary Outcome: 5-year Cumulative Incidence of Second Primary Malignancy (SPM)
Description: Second primary malignancy (SPM) is defined as the development of another new, unrelated cancer, regardless of treatment for previous malignancy attribution. The cumulative incidence of SPMs was estimated with death as a competing risk. SPMs were collected using an SAE form or MEDWATCH 3500A form, with intensity determined by using the NCI CTCAE version 4 as a guideline.
Time Frame: 5 years
Population: The analysis population is comprised of all randomized participants.
Measure: Number; unit: percentage of patients
Arm/Group | RVD Alone | RVD Plus ASCT
Number analyzed (Participants) | 357 | 365
percentage of patients | 4.9 | 6.5
Statistical Analysis 1: Comparison: RVD Alone vs RVD Plus ASCT; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.99, Log Rank; Stratified; Hazard Ratio (HR) = 1.10, 99.29% CI 2-sided [0.73 to 1.65]

10. Secondary Outcome: Median Treatment Duration
Description: Treatment duration estimated using the KM method is defined as the time from registration (C1) to the time off treatment (event) or censored at date of last treatment.
Time Frame: Up to 134 months
Population: The analysis population is comprised of all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RVD Alone | RVD Plus ASCT
Number analyzed (Participants) | 357 | 365
months | 28.2 [21.2 to 37.1] | 36.8 [29.0 to 42.2]

11. Secondary Outcome: Median Maintenance Treatment Duration
Description: Maintenance treatment duration estimated using the KM method is defined as the time from start of maintenance to the time off maintenance (event) or censored at date of last maintenance treatment.
Time Frame: Up to 128 months
Population: The analysis population is comprised of all patients that started maintenance treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RVD Alone | RVD Plus ASCT
Number analyzed (Participants) | 291 | 289
months | 36.4 [25.7 to 40.8] | 41.5 [34.0 to 47.1]

12. Secondary Outcome: Subsequent Therapy Rate
Description: Subsequent therapy rate was the percentage of participants who discontinued treatment and initiated subsequent non-protocol therapy.
Time Frame: Up to 129 months
Population: All participants off treatment per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | RVD Alone | RVD Plus ASCT
Number analyzed (Participants) | 279 | 276
Participants | 222 | 192

13. Secondary Outcome: Change From Baseline on the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACT/GOG-NTX)
Description: The FACT/GOG-NTX assessment consists of 11 questions that are all used to construct 1 subscale to summarize symptoms of peripheral neuropathy, including sensory, motor, and auditory problems and cold sensitivity. (https://www.facit.org/measures/FACT-GOG-NTX) Each question has 4 possible responses from 0 (Not at all) to 4 (Very Much) which are reverse-scored and summed. This sum is then scaled by the number of questions answered by multiplying by 11 and then dividing by the number of questions that are non-blank, in order to keep all final scores proportional to one another even if some questions are left blank. The aggregate score ranges from 0 to 44, with higher scores indicating less neurotoxicity and lower scores indicating more neurotoxicity. Change from baseline is the difference
Time Frame: Cycle 1 (Baseline), Cycle 2, Pre-Mobilization, Cycle 5 Arm A / Post Auto-HSCT Arm B, Cycle 8 Arm A /Cycle 5 Arm B, Maintenance Day 1, 2 years from baseline, 3 years from baseline
Population: The analysis population is comprised of all randomized participants who completed the assessment both at baseline and at the respective timepoint on treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RVD Alone | RVD Plus ASCT
Number analyzed (Participants) | 357 | 365
units on a scale
  Cycle 2: number analyzed (Participants) | 255 | 271
  Cycle 2 | -1.8 (4.8) | -1.3 (5.0)
  Pre-Mobilization: number analyzed (Participants) | 209 | 206
  Pre-Mobilization | -3.9 (6.9) | -3.5 (7.4)
  Cycle 5 Arm A / Post Auto-HSCT Arm B: number analyzed (Participants) | 235 | 151
  Cycle 5 Arm A / Post Auto-HSCT Arm B | -4.4 (6.5) | -4.4 (7.5)
  Cycle 8 Arm A /Cycle 5 Arm B: number analyzed (Participants) | 212 | 203
  Cycle 8 Arm A /Cycle 5 Arm B | -4.7 (6.7) | -2.5 (6.5)
  Maintenance Day 1: number analyzed (Participants) | 164 | 166
  Maintenance Day 1 | -3.7 (6.9) | -2.3 (6.4)
  2 years from baseline: number analyzed (Participants) | 99 | 118
  2 years from baseline | -4.9 (6.8) | -2.6 (6.1)
  3 years from baseline: number analyzed (Participants) | 85 | 93
  3 years from baseline | -4.6 (7.4) | -3.2 (7.2)

14. Secondary Outcome: Change From Baseline on the European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire Core 30 (EORTC QLQ-C30): Global Health Status/Quality of Life (QoL) Sub-scale
Description: The EORTC QLQ-C30 assessment consists of 30 questions that are used to construct 15 distinct sub-scales (five function scales, nine symptom scales, and a global health status/QoL scale). The global health status/QoL scale is comprised of two questions each with a range of 6 (1=Very Poor to 7=Excellent). Scores on all sub-scales range from 0 to 100 after linear transformation of the raw scores, with higher scores representing better global health status and quality of life.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RVD Alone | RVD Plus ASCT
Number analyzed (Participants) | 357 | 365
units on a scale
  Cycle 2: number analyzed (Participants) | 257 | 282
  Cycle 2 | 0.1 (20.8) | 4.3 (21.8)
  Pre-Mobilization: number analyzed (Participants) | 230 | 234
  Pre-Mobilization | 0.4 (21.7) | 4.4 (23.8)
  Cycle 5 Arm A / Post Auto-HSCT Arm B: number analyzed (Participants) | 239 | 170
  Cycle 5 Arm A / Post Auto-HSCT Arm B | 3.0 (24.8) | -11.1 (28.9)
  Cycle 8 Arm A /Cycle 5 Arm B: number analyzed (Participants) | 224 | 206
  Cycle 8 Arm A /Cycle 5 Arm B | 1.2 (23.5) | 8.3 (25.2)
  Maintenance Day 1: number analyzed (Participants) | 186 | 190
  Maintenance Day 1 | 5.3 (23.0) | 9.9 (23.6)
  2 years from baseline: number analyzed (Participants) | 107 | 127
  2 years from baseline | 5.1 (22.4) | 11.1 (26.0)
  3 years from baseline: number analyzed (Participants) | 89 | 98
  3 years from baseline | 3.5 (23.6) | 12.7 (27.4)

15. Secondary Outcome: Quality-Adjusted Life Years (QALYs)
Description: QALYs were estimated with a model beginning at initiation of first-line therapy by arm. A lifetime horizon, as well as subsequent lines of therapy, was examined using open-source Amua 0.3.0 software. Base case analysis was performed using 10,000 first-order Monte Carlo simulations. Conditional probabilities were extracted from Kaplan-Meier curves from pivotal clinical trials using WebPlotDigitizer. Costs were estimated from RED BOOK and DFCI charge reporting in US Dollars ($) after inflation adjustment to 2022 and 3% discounting, and QALYs effects were measured using EQ-5D data from Hatswell et al.
Time Frame: Maximum observation of survival for this study cohort was 129.4 months.
Measure: Mean (Standard Deviation); unit: years gained
Arm/Group | RVD Alone | RVD Plus ASCT
Number analyzed (Participants) | 357 | 365
years gained | 5.67 (3.52) | 6.10 (3.59)

16. Post Hoc Outcome: Next Generation Sequencing (NGS) Minimal Residual Disease Negative (MRD-) Rate at Maintenance Start
Description: Bone marrow aspirate samples were obtained from patients prior to the start of lenalidomide maintenance. NGS MRD- rate is the percentage of evaluable participants with MRD level of <1 x 10-5 (indicating detection of 1 malignant plasma cell in 100,000 bone marrow cells) using the validated, US Food and Drug Administration approved clonoSEQ® NGS platform (Adaptive Biotechnologies) with a minimum sensitivity of 1 x 10-5.
Time Frame: Maintenance treatment occurred after induction, up to 11.5 months.
Population: The analysis population is comprised of the participants with evaluable samples at baseline and start of maintenance.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RVD Alone | RVD Plus ASCT
Number analyzed (Participants) | 108 | 90
percentage of participants | 39.8 [30.5 to 49.7] | 54.4 [43.6 to 65.0]
Statistical Analysis 1: Comparison: RVD Alone vs RVD Plus ASCT; Test type: Superiority; Odds Ratio (OR) = 0.55, 95% CI 2-sided [0.30 to 1.01]

17. Post Hoc Outcome: Median Event Free Survival (EFS)
Description: EFS was estimated using the KM method and defined as the time from randomization to the earliest of IMWG disease progression, death, or initiation of non-protocol therapy (events); patients were censored date of last disease evaluation.
Time Frame: Assessed up to approximately 130 months.
Population: The analysis population is comprised of all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RVD Alone | RVD Plus ASCT
Number analyzed (Participants) | 357 | 365
months | 32.0 [23.5 to 42.0] | 47.3 [41.3 to 55.5]

ADVERSE EVENTS:
Time Frame: Assessed throughout the treatment period, from time of first dose and up to day 30 post-treatment. Maximum treatment duration was 133.5 months in this study cohort.
Description: Serious AEs were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv4. This is not the same definition of SAE per protocol but parallels the publication. Other AEs were defined as events with treatment-attribution of possible, probable or definite and grades 1 or 2 per CTCAEv4. Maximum grade toxicity by type was then calculated. No further data is available to specify classification of other beyond the general term.
Groups:
- RVD Cycle 1 Only: RVD cycle duration=21 days R: 25 mg oral on days 1-14 V: 1.3 mg per square meter of body surface area IV or subcutaneous on days 1, 4, 8, and 11 D: 20 mg oral (cycles 1) on days 1, 2, 4, 5, 8, 9, 11, and 12
Arm/Group | RVD Alone | RVD Plus ASCT | RVD Cycle 1 Only
All-Cause Mortality (participants affected / at risk) | 89/357 | 88/365 | 1/7
Serious Adverse Events (participants affected / at risk) | 279/357 | 344/365 | 4/7
Other Adverse Events (participants affected / at risk) | 343/357 | 345/365 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RVD Alone (N=357) | RVD Plus ASCT (N=365) | RVD Cycle 1 Only (N=7)
Anemia (Blood and lymphatic system disorders) | 65 | 108 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 15 | 33 | 0
Leukocytosis (Blood and lymphatic system disorders) | 2 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 70 | 145 | 1
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 32 | 37 | 0
Neutropenia (Blood and lymphatic system disorders) | 152 | 315 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 9 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 71 | 302 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1
Acute heart failure (Cardiac disorders) | 0 | 1 | 0
Acute pericarditis (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0
atrial flutter (Cardiac disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Conduction disorder (Cardiac disorders) | 0 | 1 | 0
Congestive heart failure (Cardiac disorders) | 1 | 3 | 0
Heart block (Cardiac disorders) | 1 | 0 | 0
Heart failure (Cardiac disorders) | 1 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 2 | 0
Paroxysmal atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0
Retinal vascular disorder (Eye disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Acute pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 3 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 0
Diarrhea (Gastrointestinal disorders) | 15 | 18 | 0
Dysphasia (Gastrointestinal disorders) | 1 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 10 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal bleed (Gastrointestinal disorders) | 2 | 2 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 2 | 1 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Mucositis (Gastrointestinal disorders) | 19 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 24 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0
Oedema uvula (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 13 | 0 | 0
Typhlitis (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 11 | 0
Chest pain (General disorders) | 3 | 0 | 0
Edema (General disorders) | 5 | 5 | 0
Edema NOS (General disorders) | 2 | 0 | 0
Fatigue (General disorders) | 10 | 22 | 0
Fever (General disorders) | 7 | 19 | 0
Malaise (General disorders) | 1 | 0 | 0
Mucositis (General disorders) | 6 | 0 | 0
Pain (General disorders) | 2 | 5 | 0
Pain NOS (General disorders) | 0 | 1 | 0
Physical deconditioning (General disorders) | 1 | 0 | 0
Sternal pain (General disorders) | 1 | 0 | 0
Sudden death (General disorders) | 1 | 0 | 0
Weakness (General disorders) | 2 | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 0
Gallbladder inflammation (Hepatobiliary disorders) | 1 | 0 | 0
Hyperbilirubinemia (Hepatobiliary disorders) | 1 | 0 | 0
Graft versus host disease (Immune system disorders) | 1 | 0 | 0
Abcess (Infections and infestations) | 2 | 0 | 0
Abdominal abscess (Infections and infestations) | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 0
Bacteremia (Infections and infestations) | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0
Breast cellulitis (Infections and infestations) | 1 | 0 | 0
Catheter infection (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 2 | 0
Clostridium difficile infection (Infections and infestations) | 3 | 0 | 0
Empyema (Infections and infestations) | 1 | 0 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0
Escherichia coli infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 2 | 0
Infection NOS (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 2 | 4 | 0
Kidney infection (Infections and infestations) | 1 | 0 | 0
Leptotrichia buccalis infection (Infections and infestations) | 1 | 0 | 0
Lip infection (Infections and infestations) | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0
Necrotizing fasciitis (Infections and infestations) | 1 | 0 | 0
Nose infection NOS (Infections and infestations) | 1 | 0 | 0
Nosocomial pneumonia (Infections and infestations) | 1 | 0 | 0
Papulopustular rash (Infections and infestations) | 2 | 0 | 0
Pneumonia (Infections and infestations) | 18 | 33 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 1 | 0
Sepsis (Infections and infestations) | 3 | 8 | 0
Shingles (Infections and infestations) | 2 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 1 | 0 | 0
Stomach virus (Infections and infestations) | 1 | 0 | 0
Streptococcal bacteremia (Infections and infestations) | 2 | 0 | 0
Streptococcal infection (Infections and infestations) | 1 | 0 | 0
Thrush (Infections and infestations) | 1 | 0 | 0
Upper respiratory infection (Infections and infestations) | 1 | 9 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 0
Viral pneumonia (Infections and infestations) | 1 | 0 | 0
Viral syndrome (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural hematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Absolute lymphocyte count decreased (Investigations) | 1 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 2 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
Creatine kinase high (Investigations) | 1 | 0 | 0
Creatinine increased (Investigations) | 1 | 0 | 0
Elevated liver enzymes (Investigations) | 8 | 8 | 1
QT interval prolonged (Investigations) | 1 | 1 | 0
Weight gain (Investigations) | 1 | 1 | 0
Weight loss (Investigations) | 1 | 0 | 0
White blood cell count increased (Investigations) | 1 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 6 | 4 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 9 | 15 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 4 | 0
Hypokalemia (Metabolism and nutrition disorders) | 12 | 7 | 0
Hyponatremia (Metabolism and nutrition disorders) | 6 | 7 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 34 | 30 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0
Ache (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Pain in elbow (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in hand (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in hip (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Pain in Neck (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain joint (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rib pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Acute lymphoblastic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
Acute lymphocytic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Acute myeloid leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast ductal cancer invasive (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ductal carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 5 | 0
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 0
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Brain stem stroke (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 0
Encephalomalacia (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 3 | 0
Memory impairment (Nervous system disorders) | 0 | 2 | 0
Neuropathy (Nervous system disorders) | 3 | 7 | 0
Sensory peripheral neuropathy (Nervous system disorders) | 17 | 19 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Stroke (Nervous system disorders) | 0 | 2 | 0
Syncope (Nervous system disorders) | 8 | 7 | 0
Anxiety (Psychiatric disorders) | 0 | 4 | 0
Confusion (Psychiatric disorders) | 0 | 2 | 0
Depression (Psychiatric disorders) | 1 | 3 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0
Incontinence (Renal and urinary disorders) | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Throat pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Facial swelling (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 | 13 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Stevens Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Cholecystostomy (Surgical and medical procedures) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0
Hypertension (Vascular disorders) | 5 | 8 | 0
Hypotension (Vascular disorders) | 4 | 9 | 0
Hypotension orthostatic (Vascular disorders) | 1 | 3 | 0
Pulmonary embolism (Vascular disorders) | 5 | 8 | 0
Thromboembolic event (Vascular disorders) | 3 | 6 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | RVD Alone (N=357) | RVD Plus ASCT (N=365) | RVD Cycle 1 Only (N=7)
Abcess (Infections and infestations) | 1 | 0 | 0
Abdominal crampy pains (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 8 | 20 | 0
Abdominal distension (Gastrointestinal disorders) | 26 | 24 | 0
Abdominal infection (Infections and infestations) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal wall cyst (Gastrointestinal disorders) | 1 | 0 | 0
Abnormal bowel sounds (Gastrointestinal disorders) | 0 | 1 | 0
Abnormal sensation in ear (Ear and labyrinth disorders) | 1 | 0 | 0
Abnormal sensation of limbs (Nervous system disorders) | 1 | 0 | 0
Abnormal vision (Eye disorders) | 5 | 2 | 0
Abrasions (Injury, poisoning and procedural complications) | 0 | 2 | 0
Abscess (Infections and infestations) | 1 | 2 | 0
Abscess jaw (Infections and infestations) | 0 | 1 | 0
Abscess limb (Infections and infestations) | 1 | 1 | 0
Abscesses of skin (Infections and infestations) | 1 | 0 | 0
Absolute lymphocyte count decreased (Investigations) | 3 | 1 | 0
Absolute monocyte count decreased (Investigations) | 0 | 1 | 0
Accidental death (General disorders) | 0 | 1 | 0
Ache (Musculoskeletal and connective tissue disorders) | 4 | 5 | 0
Achilles tendon pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Achilles tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Aching joints (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Acid reflux (Gastrointestinal disorders) | 10 | 11 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 4 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 1 | 0
Acute gastroenteritis (Infections and infestations) | 0 | 1 | 0
Acute pain (General disorders) | 1 | 1 | 0
Acute pericarditis (Cardiac disorders) | 1 | 0 | 0
Acute pharyngitis (Infections and infestations) | 1 | 0 | 0
Acute renal failure (Renal and urinary disorders) | 1 | 2 | 0
Acute renal insufficiency (Renal and urinary disorders) | 7 | 10 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acute respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute vaginitis (Infections and infestations) | 1 | 0 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Adenocarcinoma of prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0
Adverse drug reaction (General disorders) | 0 | 1 | 0
Ageusia (Nervous system disorders) | 0 | 2 | 0
Aggressive reaction (Psychiatric disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 6 | 9 | 0
Alanine aminotransferase decreased (Investigations) | 0 | 1 | 0
Albumin decreased (Investigations) | 1 | 0 | 0
Alcohol intoxication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alertness decreased (Nervous system disorders) | 0 | 1 | 0
Allergic rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Allergic reaction (Immune system disorders) | 3 | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 15 | 23 | 0
Allergy (Immune system disorders) | 6 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 55 | 23 | 0
Altered mood (Psychiatric disorders) | 1 | 2 | 0
Amnesia (Nervous system disorders) | 2 | 1 | 0
Amyloid disease (Immune system disorders) | 0 | 1 | 0
Anal bleeding (Gastrointestinal disorders) | 0 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 2 | 0
Anal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Anal lesion (Gastrointestinal disorders) | 1 | 0 | 0
Anal pain (Gastrointestinal disorders) | 1 | 0 | 0
Anaphylaxis (Immune system disorders) | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 51 | 65 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Anisocoria (Eye disorders) | 1 | 0 | 0
Ankle edema (General disorders) | 7 | 17 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Ankle injury (Injury, poisoning and procedural complications) | 1 | 2 | 0
Anorectal infection (Infections and infestations) | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 59 | 78 | 0
Anxiety (Psychiatric disorders) | 57 | 71 | 1
Anxiety depression (Psychiatric disorders) | 2 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Appetite increased (Metabolism and nutrition disorders) | 3 | 2 | 0
Application site bruise (General disorders) | 1 | 2 | 0
Arm discomfort (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Arm fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 2 | 0
Arteriovenous fistula site oedema (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 34 | 55 | 0
Arthritic pains (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 6 | 2 | 0
Articular calcification (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Articular gout (Metabolism and nutrition disorders) | 0 | 1 | 0
Aspartate aminotransferase decreased (Investigations) | 3 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 5 | 4 | 0
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Asthenia (General disorders) | 1 | 3 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Astigmatism (Eye disorders) | 0 | 1 | 0
Asystole (Cardiac disorders) | 0 | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Atherosclerosis (Vascular disorders) | 0 | 1 | 0
Athlete's foot (Infections and infestations) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 5 | 5 | 0
Atrial flutter (Cardiac disorders) | 2 | 1 | 0
Atrophy skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Attentiveness decreased (Nervous system disorders) | 1 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 1 | 0
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Avascular necrosis femoral head (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Axillary abscess (Infections and infestations) | 1 | 0 | 0
Axillary lump (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back discomfort (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 2 | 0
Back muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 147 | 132 | 0
Back stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back strain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Backache (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bacteremia (Infections and infestations) | 1 | 3 | 0
Bacterial vaginosis (Infections and infestations) | 1 | 1 | 0
Baker's cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 4 | 4 | 0
Bartholin's cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 7 | 0
Bed wetting (Renal and urinary disorders) | 0 | 1 | 0
Belching (Gastrointestinal disorders) | 2 | 5 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 1 | 0
Bilirubin total (Investigations) | 0 | 1 | 0
Bilirubin total high (Investigations) | 0 | 1 | 0
Black stools (Gastrointestinal disorders) | 2 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Bladder infection (Infections and infestations) | 0 | 1 | 0
Bladder prolapse (Renal and urinary disorders) | 1 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 0 | 0
Bleeding (Vascular disorders) | 0 | 2 | 0
Bleeding from tongue (Gastrointestinal disorders) | 0 | 1 | 0
Bleeding lips (Gastrointestinal disorders) | 1 | 0 | 0
Bleeding menstrual heavy (Reproductive system and breast disorders) | 0 | 1 | 0
Bleeding nose (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0
Bleeding nose (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 0
Bleeding time abnormal (Investigations) | 0 | 1 | 0
Blepharitis (Eye disorders) | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 2 | 4 | 0
Blister of lip (Gastrointestinal disorders) | 1 | 0 | 0
Blistering of mouth (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Blood albumin (Investigations) | 1 | 0 | 0
Blood alkaline phosphatase NOS decreased (Investigations) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 17 | 13 | 0
Blood creatinine decreased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 3 | 2 | 0
Blood in stool (Gastrointestinal disorders) | 8 | 11 | 0
Blood in urine (Investigations) | 0 | 2 | 0
Blood phosphorus increased (Investigations) | 1 | 1 | 0
Blood stool (Gastrointestinal disorders) | 0 | 1 | 0
Blood urea nitrogen decreased (Investigations) | 1 | 0 | 0
Blood urea nitrogen increased (Investigations) | 1 | 1/357 | 0
Bloodshot eye (Eye disorders) | 1 | 0 | 0
Bloody semen (Reproductive system and breast disorders) | 0 | 1 | 0
Blurred vision (Eye disorders) | 67 | 41 | 0
Body odor (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Boil (Infections and infestations) | 0 | 1 | 0
Bone density decreased (Investigations) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 53 | 52 | 0
Bone spur (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bowel cramps (Gastrointestinal disorders) | 1 | 0 | 0
Bowel movement irregularity (Gastrointestinal disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 29 | 24 | 0
Brain disorder NOS (Nervous system disorders) | 0 | 1 | 0
Breast discomfort (Reproductive system and breast disorders) | 1 | 0 | 0
Breast ductal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast lump (Reproductive system and breast disorders) | 1 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 2 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 1 | 0
Breast swelling (Reproductive system and breast disorders) | 0 | 1 | 0
Breast tenderness (Reproductive system and breast disorders) | 1 | 1 | 0
Breath shortness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Breathing difficult (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Breathlessness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Brittle nails (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Broken bones (Injury, poisoning and procedural complications) | 2 | 1 | 0
Broken foot (Injury, poisoning and procedural complications) | 0 | 1 | 0
Bronchial infection (Infections and infestations) | 3 | 4 | 0
Bronchiolitis (Infections and infestations) | 0 | 1 | 0
Bronchitis acute (Infections and infestations) | 0 | 1 | 0
Bronchitis asthmatic (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Bronchitis viral (Infections and infestations) | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bruise (Injury, poisoning and procedural complications) | 0 | 2 | 0
Bruising (Injury, poisoning and procedural complications) | 18 | 31 | 0
Bruising of face (Injury, poisoning and procedural complications) | 1 | 1 | 0
Buccal ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Bug bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
BUN increased (Investigations) | 1 | 1 | 0
Burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Burn of face, unspecified degree (Injury, poisoning and procedural complications) | 0 | 1 | 0
Burning eyes (Eye disorders) | 1 | 1 | 0
Burning leg (Nervous system disorders) | 1 | 1 | 0
Burning micturition (Renal and urinary disorders) | 1 | 0 | 0
Burning sensation in abdomen (Gastrointestinal disorders) | 0 | 1 | 0
Burning tongue (Gastrointestinal disorders) | 0 | 2 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Calcium ionized (Investigations) | 0 | 2 | 0
Calcium low (Investigations) | 0 | 1 | 0
Calf pain (Musculoskeletal and connective tissue disorders) | 2 | 9 | 0
Canker sore lip (Gastrointestinal disorders) | 1 | 0 | 0
Canker sores oral (Gastrointestinal disorders) | 3 | 3 | 0
Carbon monoxide diffusing capacity decreased (Investigations) | 0 | 2 | 0
Carbuncle (Infections and infestations) | 0 | 1 | 0
Carcinoma kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Cardiac disorder (Cardiac disorders) | 1 | 1 | 0
Caregiver (Social circumstances) | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 2 | 4 | 0
Cataract (Eye disorders) | 7 | 5 | 0
Catheter infection (Infections and infestations) | 3 | 3 | 0
Catheter placement (Surgical and medical procedures) | 1 | 0 | 0
Catheter site bleeding (General disorders) | 0 | 1 | 0
Catheter site bruise (General disorders) | 1 | 0 | 0
Catheter site erythema (General disorders) | 0 | 1 | 0
Catheter site pain (General disorders) | 1 | 1 | 0
Catheter site redness (General disorders) | 1 | 1 | 0
Cellulitis (Infections and infestations) | 8 | 16 | 0
Cellulitis of arm (Infections and infestations) | 0 | 1 | 0
Cellulitis of thumb (Infections and infestations) | 1 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Cervical pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Chalazion (Eye disorders) | 1 | 0 | 0
Cherry angiomas (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Chest cold (Infections and infestations) | 1 | 0 | 0
Chest discomfort (General disorders) | 3 | 5 | 0
Chest fullness (General disorders) | 0 | 1 | 0
Chest mass NOS (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 31 | 58 | 0
Chest pain (non-cardiac) (General disorders) | 2 | 4 | 0
Chest tenderness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Chest tightness (General disorders) | 1 | 7 | 0
Chest wall abscess (Infections and infestations) | 1 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Chills (General disorders) | 33 | 48 | 1
Chloride (Investigations) | 0 | 1 | 0
Chloride high (Investigations) | 0 | 1 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 6 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 2 | 0
Cholesterol high (Investigations) | 0 | 2 | 0
Chronic cholecystitis (Hepatobiliary disorders) | 2 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Chronic heartburn (Gastrointestinal disorders) | 1 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 3 | 1 | 0
Chronic lower extremity cellulitis (Infections and infestations) | 1 | 0 | 0
Chronic renal failure (Renal and urinary disorders) | 1 | 0 | 0
Circulating thrombus (Vascular disorders) | 1 | 1 | 0
Clonus (Nervous system disorders) | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 2 | 10 | 0
Cloudy urine (Renal and urinary disorders) | 1 | 0 | 0
Coccyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cognitive deterioration (Nervous system disorders) | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 5 | 6 | 1
Cold (Infections and infestations) | 38 | 41 | 0
Cold extremities (Vascular disorders) | 1 | 0 | 0
Cold feet (Vascular disorders) | 2 | 1 | 0
Cold intolerance (General disorders) | 0 | 1 | 0
Cold intolerance (General disorders) | 1 | 1 | 0
Cold sore (herpetic) (Infections and infestations) | 0 | 1 | 0
Cold sores (Infections and infestations) | 0 | 5 | 0
Colic biliary (Hepatobiliary disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 2 | 0
Collapsed vertebra (Injury, poisoning and procedural complications) | 0 | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 4 | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 5 | 0
Concentration impaired (Nervous system disorders) | 6 | 7 | 1
Conduction disorder (Cardiac disorders) | 0 | 2 | 0
Confusion (Psychiatric disorders) | 7 | 4 | 0
Congestion nasal (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Congestive heart failure (Cardiac disorders) | 1 | 3 | 0
Conjunctival injection (Eye disorders) | 2 | 0 | 0
Conjunctivitis (Eye disorders) | 14 | 14 | 0
Conjunctivitis bacterial (Infections and infestations) | 1 | 0 | 0
Conjunctivitis infective (Infections and infestations) | 1 | 0 | 0
Conjunctivitis, unspecified (Eye disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 192 | 196 | 1
Contact dermatitis (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Continuous urinary leakage (Renal and urinary disorders) | 1 | 0 | 0
Contusion of finger (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion of foot (Injury, poisoning and procedural complications) | 1 | 0 | 0
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Copper deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Coronary artery atherosclerosis (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 2 | 0
Coronavirus infection (Infections and infestations) | 4 | 4 | 0
Coronavirus test positive (Investigations) | 1 | 0 | 0
Correction hammer toe (Surgical and medical procedures) | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 118 | 141 | 1
Cough nonproductive (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 0
CPK increase (Investigations) | 0 | 1 | 0
Crackling jaw (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Cramps (Musculoskeletal and connective tissue disorders) | 44 | 47 | 0
Cramps in the calves (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Creatine urine increased (Investigations) | 0 | 1 | 0
Creatinine increased (Investigations) | 24 | 25 | 1
Cryoglobulins (Investigations) | 1 | 0 | 0
Cushingoid (Endocrine disorders) | 2 | 0 | 0
Cyst (General disorders) | 4 | 6 | 0
Cyst removal (Surgical and medical procedures) | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 2 | 0
Cytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Darkened skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Debridement (Surgical and medical procedures) | 1 | 0 | 0
Decreased activity (Psychiatric disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 18 | 21 | 0
Decreased INR (Investigations) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 10 | 13 | 0
Deformity thorax (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Degenerative disc disease (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 15 | 32 | 0
Delayed healing of wound (General disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 2 | 0
Delusional perception (Psychiatric disorders) | 1 | 0 | 0
Demyelinating polyneuropathy (Nervous system disorders) | 0 | 1 | 0
Dental abscess (Infections and infestations) | 3 | 2 | 0
Dental caries (Gastrointestinal disorders) | 3 | 1 | 0
Dental cavity (Gastrointestinal disorders) | 1 | 0 | 0
Dental disorder NOS (Gastrointestinal disorders) | 2 | 1 | 0
Depression (Psychiatric disorders) | 38 | 54 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 4 | 0 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0
Diabetes (Metabolism and nutrition disorders) | 0 | 2 | 0
Diaphoresis (Skin and subcutaneous tissue disorders) | 9 | 7 | 0
Diaphragmatic disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 192 | 233 | 0
Difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Difficulty in walking (General disorders) | 1 | 1 | 0
Diplopia (Eye disorders) | 0 | 3 | 0
Discoloration skin (Skin and subcutaneous tissue disorders) | 1 | 6 | 0
Dislocation of wrist (Injury, poisoning and procedural complications) | 1 | 0 | 0
Disorder equilibrium (Nervous system disorders) | 1 | 0 | 0
Disorder sperm (Investigations) | 0 | 1 | 0
Disorder tendon (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Disorder urinary tract (Renal and urinary disorders) | 0 | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 2 | 0
Distress gastrointestinal (Gastrointestinal disorders) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 2 | 2 | 0
Dizziness (Nervous system disorders) | 73 | 91 | 1
Dog bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Drenching sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
DRESS syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Drowsiness (Nervous system disorders) | 5 | 3 | 0
Drug intolerance (General disorders) | 1 | 0 | 0
Dry cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 0
Dry eyes (Eye disorders) | 30 | 21 | 0
Dry heaves (Gastrointestinal disorders) | 0 | 2 | 0
Dry lips (Gastrointestinal disorders) | 0 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 34 | 30 | 0
Dry nose (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 52 | 48 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Dysesthesia (Nervous system disorders) | 3 | 5 | 0
Dysgeusia (Nervous system disorders) | 51 | 52 | 0
Dysosmia (Nervous system disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 34 | 37 | 0
Dysphasia (Gastrointestinal disorders) | 7 | 11 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 109 | 98 | 1
Dystonic reaction (Nervous system disorders) | 0 | 2 | 0
Dysuria (Renal and urinary disorders) | 7 | 12 | 0
Ear ache (Ear and labyrinth disorders) | 2 | 3 | 0
Ear congestion (Ear and labyrinth disorders) | 3 | 2 | 0
Ear discomfort (Ear and labyrinth disorders) | 2 | 2 | 0
Ear disorder (Ear and labyrinth disorders) | 1 | 2 | 0
Ear feels clogged (Ear and labyrinth disorders) | 4 | 3 | 0
Ear infection (Infections and infestations) | 8 | 5 | 0
Ear pain (Ear and labyrinth disorders) | 10 | 16 | 0
Ear ringing (Ear and labyrinth disorders) | 1 | 0 | 0
Ear swelling (Ear and labyrinth disorders) | 0 | 1 | 0
Ear wax (Ear and labyrinth disorders) | 1 | 1 | 0
Early satiety (General disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 4 | 0
Edema (General disorders) | 157 | 143 | 0
Edema arms (General disorders) | 1 | 2 | 0
Edema face (General disorders) | 7 | 4 | 0
Edema knees (General disorders) | 1 | 1 | 0
Edema legs (General disorders) | 1 | 0 | 0
Edema of eyelid (Eye disorders) | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 2 | 0
Elbow deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Electric shock sensation (Nervous system disorders) | 1 | 0 | 0
Electrocardiogram QTc interval prolonged (Investigations) | 0 | 2 | 0
Electrolyte abnormality (Metabolism and nutrition disorders) | 0 | 1 | 0
Elevated liver enzymes (Investigations) | 54 | 56 | 1
Elevated prostate specific antigen [PSA] (Investigations) | 2 | 0 | 0
Emesis (Gastrointestinal disorders) | 2 | 6 | 0
Emesis bloody (Gastrointestinal disorders) | 0 | 1 | 0
Emotional disorder (Psychiatric disorders) | 0 | 1 | 0
Emotional distress (Psychiatric disorders) | 0 | 0 | 1
Emotional instability (Psychiatric disorders) | 1 | 0 | 0
Emotional lability (Psychiatric disorders) | 2 | 0 | 0
Empyema (Infections and infestations) | 1 | 0 | 0
Enlarged prostate (Reproductive system and breast disorders) | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 2 | 0
Enterovirus infection (Infections and infestations) | 0 | 1 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 6 | 6 | 0
Epigastric hernia (Gastrointestinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 | 11 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 9 | 9 | 0
Erythema (Skin and subcutaneous tissue disorders) | 5 | 8 | 0
Erythema eyelid (Eye disorders) | 1 | 0 | 0
Erythropapular rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Esophageal pain (Gastrointestinal disorders) | 0 | 2 | 0
Esophageal stenosis (Gastrointestinal disorders) | 0 | 1 | 0
Esophageal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Esophagitis (Gastrointestinal disorders) | 4 | 24 | 0
Essential hypertension (Vascular disorders) | 0 | 1 | 0
Exacerbation of asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Exaggerated well-being (Psychiatric disorders) | 0 | 1 | 0
Excess sweating (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Excessive thirst (General disorders) | 2 | 0 | 0
Exercise EKG abnormal (Investigations) | 1 | 1 | 0
Exercise tolerance decreased (General disorders) | 2 | 0 | 0
Exertional dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0
Exposure to poison ivy (Injury, poisoning and procedural complications) | 1 | 1 | 0
Extensive rash of forearm (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
External ear infection NOS (Infections and infestations) | 1 | 0 | 0
Extravasation (General disorders) | 1 | 0 | 0
Extremities burning sensation of (Nervous system disorders) | 1 | 0 | 0
Eye allergy (Eye disorders) | 1 | 0 | 0
Eye disorder (Eye disorders) | 1 | 1 | 0
Eye edema (Eye disorders) | 4 | 3 | 0
Eye floaters (Eye disorders) | 0 | 1 | 0
Eye infection (Infections and infestations) | 9 | 4 | 0
Eye inflammation (Eye disorders) | 1 | 2 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Eye irrigation (Surgical and medical procedures) | 0 | 1 | 0
Eye irritation (Eye disorders) | 1 | 5 | 0
Eye itching (Eye disorders) | 1 | 0 | 0
Eye muscle weakness (Eye disorders) | 0 | 1 | 0
Eye pain (Eye disorders) | 10 | 5 | 0
Eye redness (Eye disorders) | 1 | 1 | 0
Eyelid abscess drainage (Surgical and medical procedures) | 0 | 2 | 0
Eyelid injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Eyelid irritation (Eye disorders) | 0 | 1 | 0
Eyelid margin crusting (Eye disorders) | 1 | 0 | 0
Eyelid twitching (Eye disorders) | 0 | 0 | 0
Eyelid twitching (Eye disorders) | 1 | 3 | 0
Eyes swollen (Eye disorders) | 1 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Face rigidity (Nervous system disorders) | 0 | 1 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 1 | 0
Facial pain (General disorders) | 2 | 2 | 0
Facial swelling (Skin and subcutaneous tissue disorders) | 2 | 3 | 0
Faint (Nervous system disorders) | 3 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 21 | 30 | 0
Fascitis plantar (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Fatigue (General disorders) | 230 | 235 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 8 | 0
Fecal incontinence (Gastrointestinal disorders) | 2 | 0 | 0
Feeling jittery (General disorders) | 1 | 0 | 0
Feeling of warmth (General disorders) | 0 | 1 | 0
Feeling strange (General disorders) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fever (General disorders) | 96 | 113 | 2
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fine motor delay (Nervous system disorders) | 0 | 1 | 0
Finger cramps (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0
Fingers stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Fingers swollen feeling of (General disorders) | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 5 | 8 | 0
Flashing lights (Eye disorders) | 0 | 2 | 0
Flatulence (Gastrointestinal disorders) | 10 | 23 | 0
Floaters (Eye disorders) | 1 | 3 | 0
Floaters in eye (Eye disorders) | 1 | 0 | 0
Flu like symptoms (General disorders) | 41 | 43 | 0
Fluid in middle ear (Ear and labyrinth disorders) | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0
Flu-like illness (General disorders) | 1 | 0 | 0
Flu-like symptoms (General disorders) | 2 | 1 | 0
Flushing (Vascular disorders) | 8 | 8 | 1
Foggy feeling in head (General disorders) | 4 | 4 | 0
Folic acid deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Folliculitis (Infections and infestations) | 5 | 15 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 0
Foot cramps (Musculoskeletal and connective tissue disorders) | 6 | 1 | 0
Foot discomfort (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Foot drop (Nervous system disorders) | 1 | 2 | 0
Foot edema (General disorders) | 4 | 5 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Foot injury (Injury, poisoning and procedural complications) | 1 | 2 | 0
Foot pain (Musculoskeletal and connective tissue disorders) | 13 | 13 | 0
Foot sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Forehead swelling (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Forgetfulness (Nervous system disorders) | 3 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fracture femur (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fracture of metacarpal bone(s) (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fracture of spine (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fracture vertebral (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fractured finger (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fractured metatarsal (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fractured radial head (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fractured ribs (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fractured thumb (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fractured toe (Injury, poisoning and procedural complications) | 1 | 2 | 0
Fractured vertebra (compression) (Injury, poisoning and procedural complications) | 1 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0
Fungal infection (Infections and infestations) | 2 | 2 | 0
Fungal rash (Infections and infestations) | 1 | 1 | 0
Gait disorder (General disorders) | 1 | 0 | 0
Gait disturbance (General disorders) | 2 | 5 | 0
Gallbladder disease (Hepatobiliary disorders) | 0 | 1 | 0
Gallbladder pain (Hepatobiliary disorders) | 0 | 2 | 0
Gallstones (Hepatobiliary disorders) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 2 | 1 | 0
Gastritis (Gastrointestinal disorders) | 4 | 2 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 4 | 9 | 0
Gastroenteritis norovirus (Infections and infestations) | 1 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 | 16 | 0
Gastrointestinal bleed (Gastrointestinal disorders) | 3 | 2 | 0
Gastrointestinal discomfort (Gastrointestinal disorders) | 10 | 11 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 3 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 1 | 0
Gastrointestinal mucositis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal symptom NOS (Gastrointestinal disorders) | 1 | 1 | 0
Gastrointestinal viral infection (Infections and infestations) | 2 | 2 | 0
Gastroparesis (Gastrointestinal disorders) | 3 | 1 | 0
Generalized illness (General disorders) | 0 | 2 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 7 | 0
Genital abrasion (Reproductive system and breast disorders) | 0 | 1 | 0
Genital herpes (Infections and infestations) | 1 | 1 | 0
Genital labial cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Genital lesion (Reproductive system and breast disorders) | 1 | 0 | 0
Genital pain (Reproductive system and breast disorders) | 0 | 1 | 0
GERD (Gastrointestinal disorders) | 13 | 17 | 0
GI infection (Infections and infestations) | 1 | 0 | 0
GI neoplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gingival hyperpigmentation (Gastrointestinal disorders) | 0 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 1 | 0
Gingivitis (Gastrointestinal disorders) | 2 | 2 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0
Glucose high (Investigations) | 0 | 1 | 0
Glucose increased (Investigations) | 1 | 0 | 0
Goose bumps (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 4 | 9 | 0
Gout flare (Metabolism and nutrition disorders) | 0 | 2 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Gouty pain (Metabolism and nutrition disorders) | 0 | 1 | 0
Graft versus host disease (Immune system disorders) | 0 | 2 | 0
Granuloma faciale (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Grinding tooth (Psychiatric disorders) | 0 | 1 | 0
Groin abscess (Infections and infestations) | 1 | 0 | 0
Groin discomfort (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 3 | 7 | 0
Gum bleeding (Gastrointestinal disorders) | 0 | 2 | 0
Gum disorder (Gastrointestinal disorders) | 1 | 2 | 0
Gum infection (Infections and infestations) | 0 | 1 | 0
Gum pain (Gastrointestinal disorders) | 0 | 1 | 0
Gum swelling (Gastrointestinal disorders) | 1 | 1 | 0
Gynecomastia (Reproductive system and breast disorders) | 2 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Hair breakage (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hair loss (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Hallucinations (Psychiatric disorders) | 0 | 2 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Hand osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Hand pain (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0
Hand swelling (General disorders) | 2 | 0 | 0
Hands weakness of (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Hashimoto's thyroiditis (Endocrine disorders) | 1 | 0 | 0
HbA1C increased (Investigations) | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Head pain (Nervous system disorders) | 0 | 1 | 0
Head tightness (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 87 | 116 | 1
Hearing disability (Social circumstances) | 1 | 2 | 0
Hearing impaired (Ear and labyrinth disorders) | 7 | 13 | 0
Heart enlarged (Cardiac disorders) | 1 | 0 | 0
Heart murmur (Investigations) | 1 | 2 | 1
Heart rate high (Investigations) | 1 | 0 | 0
Heart rate increased (Investigations) | 2 | 1 | 0
Heartburn (Gastrointestinal disorders) | 17 | 16 | 0
Heat intolerance (General disorders) | 1 | 0 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Heat sensitivity (General disorders) | 2 | 2 | 0
Heaviness in limbs (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Helicobacter pylori gastritis (Infections and infestations) | 0 | 1 | 0
Helicobacter pylori infection (Infections and infestations) | 0 | 1 | 0
Hemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hematocrit increased (Investigations) | 0 | 1 | 0
Hematoma (Vascular disorders) | 7 | 6 | 0
Hematuria (Renal and urinary disorders) | 8 | 13 | 0
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Hemorrhage oral (Gastrointestinal disorders) | 0 | 1 | 0
Hemorrhagic cystitis (Renal and urinary disorders) | 1 | 1 | 0
Hemorrhoidal bleeding (Gastrointestinal disorders) | 2 | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 8 | 5 | 0
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hepatic lesion (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatitis C (Infections and infestations) | 0 | 1 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 1 | 0 | 0
Hernia (General disorders) | 1 | 1 | 0
Hernia inguinal (Gastrointestinal disorders) | 1 | 0 | 0
Herpes labialis (Infections and infestations) | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 2 | 3 | 0
Herpes zoster (Infections and infestations) | 8 | 14 | 0
Herpes zoster multi-dermatomal (Infections and infestations) | 0 | 1 | 0
Hiatal hernia (Gastrointestinal disorders) | 0 | 3 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 14 | 18 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
High cholesterol (Investigations) | 0 | 1 | 0
Hip discomfort (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip surgery (Surgical and medical procedures) | 0 | 1 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Hives (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 14 | 14 | 0
Hordeolum (Infections and infestations) | 2 | 2 | 0
Hot feeling in hand (General disorders) | 1 | 1 | 0
Hot flashes (Vascular disorders) | 20 | 27 | 0
Human anaplasmosis (Infections and infestations) | 0 | 1 | 0
Human papilloma virus infection (Infections and infestations) | 1 | 0 | 0
Hyperactivity (Nervous system disorders) | 0 | 1 | 0
Hyperalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperbilirubinemia (Hepatobiliary disorders) | 3 | 3 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 7 | 5 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hyperchloremic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercholesterolemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 43 | 38 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 6 | 7 | 0
Hyperlipasemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperlipidemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 5 | 6 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 7 | 0
Hyperopia (Eye disorders) | 0 | 1 | 0
Hyperpigmentation skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0
Hyperpigmentation skin (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Hypersensation skin (Nervous system disorders) | 0 | 2 | 0
Hypertension (Vascular disorders) | 72 | 69 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 9 | 9 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 17 | 18 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 48 | 54 | 2
Hypogammaglobulinaemia (Immune system disorders) | 0 | 1 | 0
Hypogeusia (Nervous system disorders) | 1 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 11 | 6 | 0
Hypokalemia (Metabolism and nutrition disorders) | 85 | 92 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 34 | 36 | 0
Hyponatremia (Metabolism and nutrition disorders) | 28 | 33 | 1
Hyponatremia aggravated (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 62 | 49 | 0
Hypotension (Vascular disorders) | 30 | 47 | 1
Hypotension orthostatic (Vascular disorders) | 2 | 10 | 0
Hypotensive (Vascular disorders) | 0 | 1 | 0
Hypothermia (General disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 6 | 5 | 0
Hypouricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypovolemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 10 | 0
Ill-defined intestinal infections (Infections and infestations) | 0 | 1 | 0
Impotence (Reproductive system and breast disorders) | 1 | 0 | 0
Incontinence (Renal and urinary disorders) | 0 | 1 | 0
Increased serum creatinine (Investigations) | 0 | 1 | 0
Increased stool urgency (Gastrointestinal disorders) | 0 | 1 | 0
Increased thirst (General disorders) | 2 | 1 | 0
Increased urinary frequency (Renal and urinary disorders) | 11 | 17 | 0
Indigestion (Gastrointestinal disorders) | 0 | 4 | 0
Infected cyst (Infections and infestations) | 0 | 1 | 0
Infected finger (Infections and infestations) | 1 | 2 | 0
Infected thumb (Infections and infestations) | 1 | 0 | 0
Infected toe (Infections and infestations) | 1 | 1 | 0
Infection ingrowing toenail (Infections and infestations) | 0 | 1 | 0
Infection localised (Infections and infestations) | 0 | 1 | 0
Infection NOS (Infections and infestations) | 4 | 1 | 0
Infection staphylococcal (Infections and infestations) | 1 | 0 | 0
Inflammation (General disorders) | 0 | 1 | 0
Inflammation localized (General disorders) | 0 | 2 | 0
Influenza (Infections and infestations) | 14 | 17 | 0
Influenza B virus infection (Infections and infestations) | 0 | 1 | 0
Infusion site extravasation (General disorders) | 0 | 1 | 0
Infusion site reaction (General disorders) | 1 | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Ingrown toe nail (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 0
Injection site reaction (General disorders) | 3 | 3 | 0
Injection site tenderness (General disorders) | 1 | 0 | 0
Injury to finger NOS (Injury, poisoning and procedural complications) | 0 | 1 | 0
Injury to kidney (Renal and urinary disorders) | 1 | 1 | 0
Injury to shoulder NOS (Injury, poisoning and procedural complications) | 0 | 1 | 0
INR decreased (Investigations) | 1 | 0 | 0
INR increased (Investigations) | 3 | 0 | 0
Insect bite NOS (Injury, poisoning and procedural complications) | 2 | 2 | 0
Insomnia (Psychiatric disorders) | 136 | 126 | 0
Iron deficiency (Metabolism and nutrition disorders) | 2 | 0 | 0
Irregular menstruation (Reproductive system and breast disorders) | 1 | 1 | 0
Irritability (General disorders) | 13 | 9 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 2 | 0 | 0
Irritation gum (Gastrointestinal disorders) | 1 | 1 | 0
Irritation lips (Gastrointestinal disorders) | 0 | 1 | 0
Irritation of eyes (Eye disorders) | 1 | 0 | 0
Itchy eyes (Eye disorders) | 0 | 1 | 0
Itchy rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Itchy scalp (Skin and subcutaneous tissue disorders) | 3 | 4 | 0
Itchy throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0
Jaw bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Jaw disorder (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0
Jaw movements disturbance (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Jaw pain (Musculoskeletal and connective tissue disorders) | 17 | 10 | 0
Jitteriness (General disorders) | 5 | 0 | 0
Joint ache (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint edema (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint inflammation (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 1 | 0
Kidney pain (Renal and urinary disorders) | 1 | 0 | 0
Kidney stones (Renal and urinary disorders) | 1 | 2 | 0
Knee derangement (Injury, poisoning and procedural complications) | 0 | 1 | 0
Knee injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
Knee sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Kyphoplasty (Surgical and medical procedures) | 0 | 1 | 0
Lability emotional (Psychiatric disorders) | 4 | 3 | 0
Labyrinthine disorders (Ear and labyrinth disorders) | 1 | 0 | 0
Labyrinthitis (Infections and infestations) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 2 | 0 | 0
Laceration of arm (Injury, poisoning and procedural complications) | 0 | 1 | 0
Laceration of face (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration of finger (Injury, poisoning and procedural complications) | 1 | 1 | 0
Laceration of foot (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration of hand (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lactate dehydrogenase increased (Investigations) | 8 | 4 | 0
Laryngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Laryngitis (Infections and infestations) | 3 | 4 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lateral epicondylitis (Injury, poisoning and procedural complications) | 0 | 1 | 0
LE rash (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Left lower quadrant pain (Gastrointestinal disorders) | 0 | 1 | 0
Left otitis externa (Infections and infestations) | 0 | 1 | 0
Left upper quadrant pain (Gastrointestinal disorders) | 2 | 1 | 0
Leg cramps (Musculoskeletal and connective tissue disorders) | 10 | 13 | 0
Leg edema (General disorders) | 1 | 1 | 0
Leg injury (Injury, poisoning and procedural complications) | 0 | 2 | 0
Leg ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Lethargy (Nervous system disorders) | 7 | 9 | 0
Leukocyte count NOS (Investigations) | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 4 | 0
Leukopenia (Blood and lymphatic system disorders) | 50 | 67 | 1
Libido decreased (Psychiatric disorders) | 3 | 5 | 0
Light headedness (Nervous system disorders) | 23 | 24 | 0
Light sensitivity to eye (Eye disorders) | 1 | 0 | 0
Light-headed (Nervous system disorders) | 0 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Limbs stiffness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Lip basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lip infection (Infections and infestations) | 1 | 1 | 0
Lip injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lip sore (Gastrointestinal disorders) | 1 | 0 | 0
Lip ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Lipase increased (Investigations) | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0
Liver function test abnormal (Investigations) | 5 | 10 | 0
Localised muscle pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Localized rash (Skin and subcutaneous tissue disorders) | 1 | 5 | 0
Localized tingling (Nervous system disorders) | 0 | 1 | 0
Loose motions (Gastrointestinal disorders) | 1 | 0 | 0
Loose stools (Gastrointestinal disorders) | 8 | 19 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0
Loss of eyelashes (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Lower abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Lower extremities weakness of (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lower urinary tract symptoms (Renal and urinary disorders) | 0 | 1 | 0
Lumbar disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Lumbar pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lung nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
Lyme disease (Infections and infestations) | 3 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 1 | 1 | 0
Lymph node palpable (Investigations) | 1 | 0 | 0
Lymph nodes enlarged (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0 | 0
Lymphedema (Vascular disorders) | 1 | 0 | 0
Lymphocytes (Investigations) | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 32 | 25 | 0
Macroglossia (Congenital, familial and genetic disorders) | 0 | 1 | 0
Macular hole (Eye disorders) | 0 | 1 | 0
Magnesium increased (Investigations) | 0 | 1 | 0
Malaise (General disorders) | 26 | 20 | 0
Malar rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 2 | 0
Mania (Psychiatric disorders) | 0 | 1 | 0
Mass (General disorders) | 0 | 1 | 0
Mean cell volume low (Investigations) | 1 | 0 | 0
Melanocytic nevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
Melena (Gastrointestinal disorders) | 2 | 0 | 0
Memory impairment (Nervous system disorders) | 25 | 27 | 0
Memory loss transient (Nervous system disorders) | 1 | 0 | 0
Meniscus rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Mental concentration decreased (Nervous system disorders) | 2 | 4 | 0
Mental disorder NOS (Psychiatric disorders) | 2 | 1 | 0
Mental distress (Psychiatric disorders) | 0 | 2 | 0
Mental impairment (Nervous system disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 2 | 0
Micturition burning (Renal and urinary disorders) | 0 | 3 | 0
Migraine (Nervous system disorders) | 4 | 7 | 0
Mitral regurgitation (Cardiac disorders) | 0 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Mobitz type I (Cardiac disorders) | 0 | 1 | 0
Mood change (Psychiatric disorders) | 1 | 3 | 0
Morton's neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Motion sickness (Ear and labyrinth disorders) | 0 | 1 | 0
Mouth cyst (Gastrointestinal disorders) | 1 | 0 | 0
Mouth injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Mucosal infection (Infections and infestations) | 1 | 1 | 0
Mucositis (Gastrointestinal disorders) | 22 | 91 | 0
Mucus from eyes (Eye disorders) | 1 | 0 | 0
Multiple allergies (Immune system disorders) | 0 | 1 | 0
Muscle cramps (Musculoskeletal and connective tissue disorders) | 38 | 30 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasm (Musculoskeletal and connective tissue disorders) | 6 | 12 | 0
Muscle strain (Injury, poisoning and procedural complications) | 3 | 1 | 0
Muscle swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle tension (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle weakness (Musculoskeletal and connective tissue disorders) | 13 | 23 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 51 | 50 | 0
Mycosis (Infections and infestations) | 1 | 0 | 0
Nail discoloration (Skin and subcutaneous tissue disorders) | 4 | 4 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Nail fungal infection NOS (Infections and infestations) | 2 | 0 | 0
Nail infection (Infections and infestations) | 1 | 1 | 0
Nasal burning (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 52 | 59 | 0
Nasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Nasal mucosal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal sinus drainage (Surgical and medical procedures) | 4 | 4 | 0
Nausea (Gastrointestinal disorders) | 155 | 218 | 2
Neck discomfort (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Neck edema (General disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 26 | 37 | 0
Neck rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Neck strain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Neck swelling (General disorders) | 1 | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Nerve compression (Nervous system disorders) | 1 | 1 | 0
Nerve pain (Nervous system disorders) | 1 | 2 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 6 | 3 | 0
Neuropathy (Nervous system disorders) | 52 | 40 | 0
Neutropenia (Blood and lymphatic system disorders) | 62 | 95 | 1
Nevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 15 | 24 | 0
Nightmares (Psychiatric disorders) | 1 | 0 | 0
Nipple discharge (Reproductive system and breast disorders) | 1 | 0 | 0
Nipple tenderness (Reproductive system and breast disorders) | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 9 | 11 | 0
Nodular fasciitis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Nodule (General disorders) | 1 | 2 | 0
Nodule on extremity (General disorders) | 0 | 1 | 0
Non ST segment elevation myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 8 | 0
Norovirus test positive (Investigations) | 1 | 2 | 0
Nose infection NOS (Infections and infestations) | 1 | 0 | 0
Nose injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Nosocomial pneumonia (Infections and infestations) | 0 | 1 | 0
Numbness (Nervous system disorders) | 6 | 7 | 0
Numbness facial (Nervous system disorders) | 1 | 2 | 0
Numbness in face (Nervous system disorders) | 0 | 1 | 0
Numbness lips (Gastrointestinal disorders) | 1 | 0 | 0
Numbness localised (Nervous system disorders) | 0 | 1 | 0
Numbness localised (Nervous system disorders) | 1 | 0 | 0
Numbness of extremities (Nervous system disorders) | 8 | 15 | 0
Numbness of tongue (Gastrointestinal disorders) | 0 | 1 | 0
Numbness of upper arm (Nervous system disorders) | 1 | 0 | 1
Obstructive sleep apnea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oedema trunk (General disorders) | 1 | 0 | 0
Optic neuritis (Nervous system disorders) | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 7 | 12 | 0
Oral dysesthesia (Gastrointestinal disorders) | 1 | 0 | 0
Oral hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Oral infection (Infections and infestations) | 1 | 0 | 0
Oral intake reduced (Metabolism and nutrition disorders) | 1 | 1 | 0
Oral lesion (Gastrointestinal disorders) | 0 | 1 | 0
Oral mucosal erythema (Gastrointestinal disorders) | 0 | 1 | 0
oral pain (Gastrointestinal disorders) | 6 | 6 | 0
Orbital cellulitis (Infections and infestations) | 1 | 1 | 0
Organizing pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Orthopnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Orthostatic hypertension (Vascular disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 12 | 6 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Otitis (Infections and infestations) | 2 | 2 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 6 | 0
Otitis media (Infections and infestations) | 3 | 0 | 0
Overgrowth bacterial (Infections and infestations) | 0 | 1 | 0
Pain (General disorders) | 109 | 105 | 1
Pain abdominal (Gastrointestinal disorders) | 1 | 0 | 0
Pain back (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain bone (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain flank (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Pain foot (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Pain foot (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain groin (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in ankle (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0
Pain in arm (Musculoskeletal and connective tissue disorders) | 14 | 12 | 0
Pain in elbow (Musculoskeletal and connective tissue disorders) | 10 | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 36 | 33 | 0
Pain in face (General disorders) | 1 | 0 | 0
Pain in fingers (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in hand (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Pain in hip (Musculoskeletal and connective tissue disorders) | 48 | 32 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in joint (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in leg (Musculoskeletal and connective tissue disorders) | 20 | 21 | 0
Pain in legs (Musculoskeletal and connective tissue disorders) | 17 | 24 | 0
Pain in muscle (Musculoskeletal and connective tissue disorders) | 12 | 13 | 0
Pain in Neck (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Pain in shoulder (Musculoskeletal and connective tissue disorders) | 40 | 49 | 0
Pain in tongue (Gastrointestinal disorders) | 2 | 0 | 0
Pain in tooth (Gastrointestinal disorders) | 14 | 15 | 0
Pain in upper extremities (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Pain in wrist (Musculoskeletal and connective tissue disorders) | 4 | 8 | 0
Pain joint (Musculoskeletal and connective tissue disorders) | 9 | 12 | 0
Pain knee (Musculoskeletal and connective tissue disorders) | 19 | 17 | 0
Pain localized (General disorders) | 0 | 3 | 0
Pain lower ribs (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Pain mouth (Gastrointestinal disorders) | 1 | 0 | 0
Pain NOS (General disorders) | 8 | 13 | 0
Pain sacroiliac (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Painful L arm (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Painful urination (Renal and urinary disorders) | 1 | 1 | 0
Pains in legs (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pallor (Vascular disorders) | 1 | 2 | 0
Palmar erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Palpitations (Cardiac disorders) | 9 | 11 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 3 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 3 | 0
Panic attack (Psychiatric disorders) | 2 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Papulopustular rash (Infections and infestations) | 6 | 7 | 0
Paraesthesia hand (Nervous system disorders) | 1 | 0 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 0
Paresthesia (Nervous system disorders) | 54 | 42 | 0
Paresthesia hand (Nervous system disorders) | 1 | 0 | 0
Paresthesia of genital female (Reproductive system and breast disorders) | 1 | 0 | 0
Paresthesia upper limb (Nervous system disorders) | 1 | 0 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0
Parotid gland inflammation (Gastrointestinal disorders) | 1 | 0 | 0
Parotiditis (Infections and infestations) | 0 | 1 | 0
Parotitis (Infections and infestations) | 0 | 1 | 0
Paroxysmal atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Pelvic congestion syndrome (Reproductive system and breast disorders) | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 4 | 3 | 0
Penetrating abdominal trauma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Penis injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Perforation of tympanic membrane (Ear and labyrinth disorders) | 2 | 0 | 0
Perianal bleeding (Gastrointestinal disorders) | 1 | 0 | 0
Periapical abscess without sinus (Infections and infestations) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 3 | 0
Periodontal disease (Gastrointestinal disorders) | 2 | 1 | 0
Perioral numbness (Gastrointestinal disorders) | 0 | 1 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0 | 0
Periorbital edema (Eye disorders) | 5 | 6 | 0
Perirectal abscess (Infections and infestations) | 1 | 0 | 0
Periumbilical pain (Gastrointestinal disorders) | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Peyronie's disease (Reproductive system and breast disorders) | 1 | 0 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 2 | 5 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Phlebitis superficial (Vascular disorders) | 1 | 0 | 0
Phlegm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Phosphate decreased (Investigations) | 1 | 1 | 0
Phosphorus low (Investigations) | 0 | 1 | 0
Photophobia (Eye disorders) | 1 | 3 | 0
Pinkeye (Infections and infestations) | 2 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Plantar warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Plasma cell leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pneumonia (Infections and infestations) | 38 | 58 | 0
Poison ivy rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Poison oak rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Polyp (General disorders) | 0 | 1 | 0
Polyuria (Renal and urinary disorders) | 0 | 2 | 0
Popliteal cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 1 | 4 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 8 | 20 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Premenstrual dysphoric disorder (Reproductive system and breast disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 9 | 6 | 0
Proctocolitis (Gastrointestinal disorders) | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7 | 10 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 1 | 0
Protein-calorie malnutrition (Metabolism and nutrition disorders) | 0 | 2 | 0
Proteins serum plasma low (Investigations) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 2 | 2 | 0
Prothrombin increased (Investigations) | 0 | 1 | 0
Prothrombin time increased (Investigations) | 0 | 2 | 0
Proximal myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 25 | 40 | 0
Pseudogout (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pseudoseizure (Psychiatric disorders) | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
Psoriatic arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Psychomotor development impaired (Nervous system disorders) | 1 | 0 | 0
Psychotic episode (Psychiatric disorders) | 1 | 0 | 0
PTH increased (Investigations) | 0 | 1 | 0
Pulled muscle (Injury, poisoning and procedural complications) | 0 | 2 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary embolism (Vascular disorders) | 0 | 4 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Puncture wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 3 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Pyrosis (Gastrointestinal disorders) | 1 | 0 | 0
QT interval prolonged (Investigations) | 3 | 1 | 0
Radiculitis (Nervous system disorders) | 1 | 0 | 0
Radiculopathy (Nervous system disorders) | 0 | 2 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 3 | 4 | 0
Rash face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0
Rash face (Skin and subcutaneous tissue disorders) | 3 | 4 | 0
Rash follicular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 113 | 126 | 1
Rash over arms (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 7 | 12 | 0
Rash scaly (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Reactive airways disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rectal bleeding (Gastrointestinal disorders) | 3 | 7 | 0
Rectal blood loss (Gastrointestinal disorders) | 1 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Rectal fissure (Gastrointestinal disorders) | 0 | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Rectal pain (Gastrointestinal disorders) | 1 | 6 | 0
Red eye (Eye disorders) | 1 | 0 | 0
Renal calculi (Renal and urinary disorders) | 2 | 2 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Renal disease (Renal and urinary disorders) | 1 | 0 | 0
Renal function aggravated (Renal and urinary disorders) | 0 | 1 | 0
Renal function decreased (Investigations) | 2 | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0
Renal insufficiency (Renal and urinary disorders) | 1 | 2 | 0
Renal tract inflammation (Renal and urinary disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory infection (Infections and infestations) | 2 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 3 | 1 | 0
Resting tremor (Nervous system disorders) | 0 | 1 | 0
Restless leg syndrome (Nervous system disorders) | 5 | 5 | 0
Restlessness (Psychiatric disorders) | 0 | 7 | 0
Retinal atrophy (Eye disorders) | 0 | 1 | 0
Retinal telangiectasia (Eye disorders) | 1 | 0 | 0
Retro-orbital pain (Eye disorders) | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 9 | 11 | 0
Rhinitis infective (Infections and infestations) | 0 | 1 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 19 | 21 | 0
Rhinovirus infection (Infections and infestations) | 0 | 3 | 0
Rhinovirus infection NOS (Infections and infestations) | 0 | 1 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Rib fracture (Injury, poisoning and procedural complications) | 2 | 5 | 0
Rib injury (Injury, poisoning and procedural complications) | 2 | 0 | 0
Rib pain (Musculoskeletal and connective tissue disorders) | 21 | 24 | 0
Right upper quadrant pain (Gastrointestinal disorders) | 2 | 1 | 0
Rigors (General disorders) | 0 | 2 | 0
Ringing in ears (Ear and labyrinth disorders) | 3 | 2 | 0
Ringworm NOS (Infections and infestations) | 1 | 0 | 0
Root canal procedure (Surgical and medical procedures) | 0 | 2 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 5 | 2 | 0
Rotator cuff injury (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Rotator cuff repair (Surgical and medical procedures) | 1 | 0 | 0
Rotator cuff tear (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Sacral edema (General disorders) | 1 | 0 | 0
Sacral pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Scabbing (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Scabies (Infections and infestations) | 0 | 1 | 0
Scalp disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Scalp laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Scalp pain (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Scalp plaque (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Scapula pain (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0
Sciatica (Nervous system disorders) | 1 | 2 | 0
Scleral haemorrhage (Eye disorders) | 1 | 1 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 1 | 0
Scrotal infection (Infections and infestations) | 0 | 1 | 0
Scrotal pain (Reproductive system and breast disorders) | 0 | 1 | 0
Scrotal swelling (Reproductive system and breast disorders) | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 5 | 3 | 0
Sebaceous cyst (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Seborrhea capitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Seborrheic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Seborrheic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Second rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Seizure (Nervous system disorders) | 1 | 1 | 0
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Sensation of pressure in ear (Ear and labyrinth disorders) | 2 | 1 | 0
Sensitivity of teeth (Gastrointestinal disorders) | 3 | 4 | 0
Sensory neuropathy (Nervous system disorders) | 0 | 1 | 0
Sensory peripheral neuropathy (Nervous system disorders) | 247 | 232 | 0
Sepsis (Infections and infestations) | 2 | 5 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0
Serum ferritin abnormal (Investigations) | 0 | 1 | 0
Sexual dysfunction (Reproductive system and breast disorders) | 1 | 2 | 0
SGPT increased (Investigations) | 1 | 0 | 0
Shin splints (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Shingles (Infections and infestations) | 4 | 9 | 0
Shoulder blade pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Shoulder deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 19 | 14 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 23 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 0
Sinus headache (Nervous system disorders) | 1 | 0 | 0
Sinus infection (Infections and infestations) | 5 | 12 | 0
Sinus pain (Nervous system disorders) | 6 | 3 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 9 | 0
Sinusitis (Infections and infestations) | 29 | 42 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 2 | 1 | 0
Skin biopsy (Investigations) | 0 | 1 | 0
Skin bleeding (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Skin carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Skin cold clammy (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 4 | 0 | 0
Skin dry (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 5 | 7 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin infection (Infections and infestations) | 12 | 13 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 5 | 9 | 0
Skin peeling (Skin and subcutaneous tissue disorders) | 0 | 0 | 0
Skin peeling (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Skin pigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin rash (Skin and subcutaneous tissue disorders) | 6 | 2 | 0
Skin scaly (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin seborrheic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin sensitization (Skin and subcutaneous tissue disorders) | 0 | 0 | 0
Skin sensitization (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Skin striae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin swelling (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin tear (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin tenderness (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 2 | 0
Sleep disturbance (Psychiatric disorders) | 3 | 1 | 0
Sleep walking (Psychiatric disorders) | 0 | 1 | 0
Sleepiness (Nervous system disorders) | 1 | 1 | 0
Slight temperature (General disorders) | 0 | 1 | 0
Slurred speech (Nervous system disorders) | 0 | 3 | 0
Small bowel obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Smell alteration (Nervous system disorders) | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sodium high (Investigations) | 1 | 0 | 0
Sodium low (Investigations) | 0 | 1 | 0
Soft stools (Gastrointestinal disorders) | 0 | 2 | 0
Soft tissue infection (Infections and infestations) | 0 | 1 | 0
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Solar dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0
Sore feet (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Sore mouth (Gastrointestinal disorders) | 9 | 9 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 34 | 49 | 0
Spasms (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0
Spasticity (Nervous system disorders) | 1 | 0 | 0
Specific allergy (drug) (Immune system disorders) | 0 | 1 | 0
Spider bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 2 | 3 | 0
Splinter (Injury, poisoning and procedural complications) | 1 | 0 | 0
Sporotrichosis (Infections and infestations) | 1 | 0 | 0
Spotting menstrual (Reproductive system and breast disorders) | 0 | 1 | 0
Spotting vaginal (Reproductive system and breast disorders) | 0 | 5 | 0
Sprained ankle (Injury, poisoning and procedural complications) | 0 | 2 | 0
Sputum abnormal (Investigations) | 0 | 1 | 0
Sputum bloody (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 6 | 0
Staphylococcal infection (Infections and infestations) | 0 | 2 | 0
Sternal pain (General disorders) | 0 | 0 | 0
Sternal pain (General disorders) | 2 | 7 | 0
Sticky feeling in eyes (Eye disorders) | 0 | 1 | 0
Stiff back (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Stiff neck (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Stiffness (Musculoskeletal and connective tissue disorders) | 5 | 9 | 0
Stiffness hip (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Stiffness shoulder (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Stomach ache (Gastrointestinal disorders) | 0 | 1 | 0
Stomach flu (Infections and infestations) | 4 | 2 | 0
Stomach pain (Gastrointestinal disorders) | 69 | 72 | 0
Stomach virus (Infections and infestations) | 1 | 1 | 0
Stomachache (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Strain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Streptococcal sore throat (Infections and infestations) | 1 | 0 | 0
Stress (Psychiatric disorders) | 2 | 0 | 0
Stress fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Stroke (Nervous system disorders) | 1 | 0 | 0
Stye (Infections and infestations) | 22 | 11 | 0
Subconjunctival hemorrhage (Eye disorders) | 0 | 0 | 0
Subconjunctival hemorrhage (Eye disorders) | 1 | 1 | 0
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Subdural hematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Submaxillary gland swelling (Gastrointestinal disorders) | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 2 | 0
Sun spots (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 3 | 0 | 0
Superficial thrombophlebitis (Vascular disorders) | 2 | 1 | 0
Superficial thrombosis of veins (Vascular disorders) | 1 | 0 | 0
Suprapubic pain (General disorders) | 0 | 1 | 0
Supraspinatus syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Surgical procedure (Surgical and medical procedures) | 1 | 0 | 0
Suture insertion (Surgical and medical procedures) | 1 | 0 | 0
Swallowing difficult (Gastrointestinal disorders) | 0 | 3 | 0
Sweating (Skin and subcutaneous tissue disorders) | 0 | 0 | 0
Sweating (Skin and subcutaneous tissue disorders) | 6 | 10 | 0
Sweating and Sweaty (Skin and subcutaneous tissue disorders) | 0 | 0 | 0
Sweating and Sweaty (Skin and subcutaneous tissue disorders) | 4 | 9 | 0
Sweating increased (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Swelling of knees (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Swelling of L knee (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Swelling of R knee (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Swelling of tongue (Gastrointestinal disorders) | 1 | 0 | 0
Swollen glands (Blood and lymphatic system disorders) | 1 | 0 | 0
Swollen lymph nodes (Blood and lymphatic system disorders) | 0 | 4 | 0
Swollen thumb (General disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 8 | 13 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Syphilis (Infections and infestations) | 0 | 1 | 0
Systolic murmur (Investigations) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 10 | 28 | 0
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Taste alteration (Nervous system disorders) | 3 | 12 | 0
Taste diminished (Nervous system disorders) | 0 | 1 | 0
Teary eyes (Eye disorders) | 5 | 9 | 1
Temporomandibular joint disorder (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Tenderness (Musculoskeletal and connective tissue disorders) | 1 | 5 | 0
Tendinitis (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Tennis elbow (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tension headaches (Nervous system disorders) | 1 | 0 | 0
Testicular disorder (Reproductive system and breast disorders) | 1 | 1 | 0
Testicular edema (Reproductive system and breast disorders) | 1 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 2 | 0 | 0
Testis discomfort (Reproductive system and breast disorders) | 1 | 0 | 0
Testosterone low (Investigations) | 0 | 3 | 0
Thirst (General disorders) | 1 | 2 | 0
Thoracic spondylosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Throat infection (Infections and infestations) | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Throat pain (Respiratory, thoracic and mediastinal disorders) | 3 | 10 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 40 | 84 | 2
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Thromboembolic event (Vascular disorders) | 9 | 21 | 0
Thrombosis (Vascular disorders) | 1 | 3 | 0
Thrush (Infections and infestations) | 6 | 13 | 0
Thyroid cyst (Endocrine disorders) | 0 | 1 | 0
Thyroid hot nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Thyroid nodular (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Thyroid nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0
Thyroid nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0
Thyroid stimulating hormone increased (Investigations) | 0 | 1 | 0
Tibia pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0
Tick bite (Injury, poisoning and procedural complications) | 3 | 3 | 0
Tightness of back muscles (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tinea capitis (Infections and infestations) | 0 | 1 | 0
Tinea corporis (Infections and infestations) | 0 | 1 | 0
Tinea cruris (Infections and infestations) | 0 | 1 | 0
Tinea pedis (Infections and infestations) | 0 | 2 | 0
Tingling lips (Gastrointestinal disorders) | 1 | 0 | 0
Tingling skin (Nervous system disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 18 | 14 | 0
Tired eyes (Eye disorders) | 0 | 1 | 0
Toe injury (Injury, poisoning and procedural complications) | 2 | 2 | 0
Tongue blistering (Gastrointestinal disorders) | 0 | 1 | 0
Tongue disorder (Gastrointestinal disorders) | 4 | 0 | 0
Tongue edema (Gastrointestinal disorders) | 0 | 1 | 0
Tongue infection (Infections and infestations) | 1 | 1 | 0
Tongue injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
Tongue swelling non-specific (Gastrointestinal disorders) | 0 | 1 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 3 | 4 | 0
Tooth ache (Gastrointestinal disorders) | 1 | 2 | 0
Tooth extraction (Surgical and medical procedures) | 4 | 3 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 3 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0
Tooth infection (Infections and infestations) | 9 | 8 | 0
Tooth injury (Injury, poisoning and procedural complications) | 0 | 0 | 0
Tooth injury (Injury, poisoning and procedural complications) | 3 | 3 | 0
Torn muscle (Injury, poisoning and procedural complications) | 1 | 0 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tracheal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Transaminases increased (Investigations) | 2 | 1 | 0
Transaminitis (Investigations) | 3 | 6 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Transient insomnia (Psychiatric disorders) | 1 | 1 | 0
Transient ischemic attacks (Nervous system disorders) | 0 | 2 | 0
Tremor (Nervous system disorders) | 34 | 32 | 0
Trigeminy (Cardiac disorders) | 0 | 1 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Triglycerides (Investigations) | 0 | 1 | 0
Trochanteric bursitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
TSH increased (Investigations) | 0 | 1 | 0
Twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Ulcer mouth (Gastrointestinal disorders) | 2 | 4 | 0
Ulceration of intestine (Gastrointestinal disorders) | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 2 | 0 | 0
Uncontrolled hypertension (Vascular disorders) | 1 | 0 | 0
Unilateral leg pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 0
Unspecified disease of hair and hair follicles (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Upper back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 165 | 180 | 0
Upset stomach (Gastrointestinal disorders) | 6 | 7 | 0
Urethral burning on micturition (Renal and urinary disorders) | 0 | 1 | 0
Urgency urination (Renal and urinary disorders) | 0 | 1 | 0
Uric acid decreased (Investigations) | 2 | 0 | 0
Uric acid high (Investigations) | 1 | 0 | 0
Uric acid increased (Investigations) | 2 | 3 | 0
Urinary hesitancy (Renal and urinary disorders) | 0 | 3 | 0
Urinary incontinence (Renal and urinary disorders) | 6 | 3 | 0
Urinary infection (Infections and infestations) | 1 | 0 | 0
Urinary obstruction unspecified (Renal and urinary disorders) | 1 | 0 | 0
Urinary output diminished (Investigations) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 3 | 3 | 0
Urinary tract infection (Infections and infestations) | 26 | 32 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 2 | 0
Urinary urgency (Renal and urinary disorders) | 2 | 8 | 0
Urination difficulty (Renal and urinary disorders) | 2 | 2 | 0
Urination frequency of (Renal and urinary disorders) | 2 | 2 | 0
Urination pain (Renal and urinary disorders) | 1 | 0 | 0
Urine color abnormal (Investigations) | 0 | 1 | 0
Urine discoloration (Renal and urinary disorders) | 1 | 0 | 0
Urine output decreased (Investigations) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Urticaria localised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Uterine bleeding (Reproductive system and breast disorders) | 0 | 1 | 0
Uterine fibroid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Uveitis (Eye disorders) | 1 | 0 | 0
Uvulitis (Gastrointestinal disorders) | 1 | 0 | 0
Vaginal bleeding (Reproductive system and breast disorders) | 4 | 3 | 0
Vaginal cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal discomfort (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal dryness (Reproductive system and breast disorders) | 2 | 2 | 0
Vaginal infection (Infections and infestations) | 2 | 5 | 0
Vaginal inflammation (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal irritation (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal itching (Reproductive system and breast disorders) | 0 | 6 | 0
Vaginal lesion (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal pain (Reproductive system and breast disorders) | 1 | 2 | 0
Varicose vein (Vascular disorders) | 0 | 1 | 0
Varicosity (Vascular disorders) | 1 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Venipuncture site pain (General disorders) | 1 | 0 | 0
Venous ulcer NOS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Verruca (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 17 | 10 | 0
Vestibular disorder (Ear and labyrinth disorders) | 1 | 0 | 0
Viral gastroenteritis (Infections and infestations) | 2 | 2 | 0
Viral infection (Infections and infestations) | 6 | 7 | 0
Viral laryngitis (Infections and infestations) | 1 | 0 | 0
Viral meningitis (Infections and infestations) | 0 | 1 | 0
Viral pharyngitis (Infections and infestations) | 0 | 1 | 0
Viral pneumonia (Infections and infestations) | 0 | 3 | 0
Viral syndrome (Infections and infestations) | 1 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Vision abnormal (Eye disorders) | 2 | 4 | 0
Vision double (Eye disorders) | 1 | 0 | 0
Vision loss (Eye disorders) | 1 | 0 | 0
Visual discomfort (Eye disorders) | 1 | 0 | 0
Visual disturbances (Eye disorders) | 1 | 1 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 1 | 0
Vitamin D decreased (Investigations) | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 4 | 12 | 0
Vitreous detachment (Eye disorders) | 0 | 1 | 0
Vivid dreams (Psychiatric disorders) | 1 | 0 | 0
Vocal cord nodule (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 64 | 127 | 2
Vulval lesion (Reproductive system and breast disorders) | 0 | 1 | 0
Vulvovaginal atrophy (Reproductive system and breast disorders) | 1 | 0 | 0
Wart (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Wax in ear (Ear and labyrinth disorders) | 1 | 0 | 0
Weakness (General disorders) | 13 | 21 | 0
Weakness left or right side (Nervous system disorders) | 0 | 1 | 0
Weakness of arms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Weight gain (Investigations) | 30 | 21 | 0
Weight loss (Investigations) | 34 | 28 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 9 | 14 | 0
White blood cell count increased (Investigations) | 0 | 2 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 2 | 0
Wound breakdown (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound drainage (Surgical and medical procedures) | 2 | 0 | 0
Wound infection (Infections and infestations) | 3 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Yeast infection (Infections and infestations) | 3 | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-07-12): https://cdn.clinicaltrials.gov/large-docs/62/NCT01208662/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-12): https://cdn.clinicaltrials.gov/large-docs/62/NCT01208662/SAP_001.pdf